#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# **Clinical Study Protocol**

A Phase 2, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of VX-440 Combination Therapy in Subjects Aged 12 Years and Older With Cystic Fibrosis

Vertex Study Number: VX15-440-101

EudraCT Number: 2016-000454-36

**Date of Protocol:** 16 September 2016 (Version 2.0)

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### CONFIDENTIAL

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

#### 2 PROTOCOL SYNOPSIS

Title A Phase 2, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of VX-440 Combination Therapy in Subjects Aged 12 Years and Older With

Cystic Fibrosis

Brief Title A Study Evaluating the Safety and Efficacy of VX-440 Combination Therapy in

Subjects With Cystic Fibrosis

### Clinical Phase and Phase 2 safety and efficacy Clinical Study Type

#### Objectives **Primary Objectives**

- To evaluate the safety and tolerability of VX-440 in triple combination with tezacaftor (TEZ) and ivacaftor (IVA)
- To evaluate the efficacy of VX-440 in triple combination with TEZ and IVA

#### Secondary Objectives

- To evaluate the pharmacodynamic (PD) effect of VX-440 in triple combination with TEZ and IVA on sweat chloride concentrations
- To evaluate the pharmacokinetics (PK) of VX-440 when administered in triple combination with TEZ and IVA
- To evaluate the PK of TEZ, IVA, and their respective metabolites when administered with VX-440

### **Endpoints Primary Endpoints**

- · Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values, standard 12-lead electrocardiograms (ECGs), vital signs, and pulse oximetry
- Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline through Day 29 (Parts 1 and 2)

#### Secondary Endpoints

- Absolute change in sweat chloride concentrations from baseline through Day 29 (Parts 1 and 2)
- Relative change in ppFEV<sub>1</sub> from baseline through Day 29 (Parts 1 and 2)

- Absolute change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory domain score from baseline at Day 29 (Parts 1 and 2)
- PK parameters of VX-440, TEZ, M1-TEZ, IVA, and M1-IVA

Number of Subjects

Approximately 198 subjects will be randomized: approximately 42 subjects in Part 1,

approximately 24 subjects in Part 2

**Study Population** Male and female subjects with cystic fibrosis (CF)

Part 1: F508del/minimal function (MF) genotype, 18 years of age or older

Part 2: F508del/F508del genotype, 18 years of age or older

Investigational Drug Active substance: VX-440

Activity: CF transmembrane conductance regulatory (CFTR) corrector (increased

chloride ion [Cl] secretion)

Strength and route of administration: 200-mg tablet for oral administration

Active substance: TEZ (tezacaftor; VX-661) and IVA (ivacaftor; VX-770)

Activity: CFTR corrector and potentiator (increased Cl secretion)

Strength and route of administration: 100-mg TEZ/150-mg IVA fixed-dose

combination (light yellow) film-coated tablet for oral administration

Active substance: TEZ

Activity: CFTR corrector (increased Cl secretion)

Strength and route of administration: 50-mg (white) tablet for oral administration

Active substance: IVA

Activity: CFTR potentiator (increased Cl<sup>-</sup> secretion)

Strength and route of administration: 150-mg IVA (light blue) film-coated tablet for

oral administration

Active substance: not applicable

Activity: VX-440-matching placebo, TEZ/IVA-matching placebo, TEZ-matching

placebo, IVA-matching placebo

Strength and route of administration: 0-mg film-coated matching placebo tablets for

oral administration

#### Study Duration Part 1

The total study duration is approximately 12 weeks (4 weeks for the Screening Period, 4 weeks for the Treatment Period, and 4 weeks for the Safety Follow-up Period). Subjects will receive study drug for approximately 4 weeks.

#### Part 2

The total study duration is approximately 20 weeks (4 weeks for the Screening Period, 4 weeks for the Run-in Period, 4 weeks for the Treatment Period, 4 weeks for the Washout Period, and 4 weeks for the Safety Follow-up Period). Subjects will receive study drug for approximately 12 weeks (4 weeks of TEZ/IVA during the Run-in Period, 4 weeks of VX-440 or placebo + TEZ/IVA during the Treatment Period, and 4 weeks of TEZ/IVA during the Washout Period).



#### Study Design

This is a Phase 2, randomized, double-blind, placebo- and TEZ/IVA-controlled, parallel group, multicenter study. The treatment arms and doses of VX-440, TEZ, and IVA to be evaluated are shown in the table below.

Part 1 will consist of 2 cohorts: Cohort 1A and Cohort 1B. The start of dosing of Cohort 1A and Cohort 1B will be sequential. After all Cohort 1A subjects complete the Day 15 Visit, a blinded review of all available safety and PK data will be conducted by the Vertex study team and lead investigator(s). Dosing of Cohort 1B will begin after the blinded review, if supported by safety and PK data.

Part 2 will initiate after the Cohort 1A blinded review, if supported by safety and PK data.



Treatment Arms and Planned Doses by Part

| Part | Treatment Arm | VX-440 Dosage | TEZ Dosage | IVA Dosage |
|-----------|----------------|---------------|------------|-------------|
| Part 1 | TC-1A | 200 mg q12h | 100 mg qd | 150 mg q12h |
| Cohort 1A | Triple placebo | Placebo | Placebo | Placebo |
| Part 1 | TC-1B-high | 600 mg q12h | 50 mg q12h | 300 mg q12h |
| Cohort 1B | TC-1B-low | 200 mg q12h | 50 mg q12h | 150 mg q12h |
| | Triple placebo | Placebo | Placebo | Placebo |
| Part 2 | TC-2 | 600 mg q12h | 50 mg q12h | 300 mg q12h |
| | TEZ/IVA | Placebo | 100 mg qd | 150 mg q12h |

IVA: ivacaftor; q12h: every 12 hours; qd: daily; TBD: to be determined; TEZ: tezacaftor Notes: In the "TC-1B-high" and "TC-2" treatment arms, the dosage of VX-440 will be determined based on safety and PK data from Cohort 1A. The planned dose is shown, but may be reduced to 400 mg q12h

#### Schematics of the study design are shown below.

Part 1 Cohort 1A: F508del/MF (N ~ 10) Randomization: 4:1

N = 8
TC-1A
Triple placebo

4 Weeks

Part 1 Cohort 1B: F508del/MF (N ~ 32) Randomization: 2:1:1

Stratification: ppFEV1: ≥70 versus <70

| N=16 | TC-1B-high |
|-------|----------------|
| N = 8 | TC-1B-low |
| N = 8 | Triple placebo |
| | 4 Weeks |

Part 2: F508del/F508del (N ~ 24) Randomization: 3:1

Stratification: ppFEV<sub>1</sub>: ≥70 versus <70

| | Run-in Period | Treatment Period | Washout Period |
|---|---|---|---|
| N = 18 | TE 7/TV A | TC-2 (VX-440 + TEZ/IVA) | TEZ/IVA |
| N = 6 | TEZ/IVA | Placebo + TEZ/IVA | IEZ/IVA |
| | Day -28 through<br>Day -1 | , w. h | Day 29 through<br>Day 57 |



#### Assessments

**Safety:** AEs, clinical laboratory assessments, ECGs, vital signs, pulse oximetry, physical examinations (PEs), and ophthalmologic examinations

Efficacy: spirometry, height, weight, CFQ-R

PD: sweat chloride

PK: VX-440, TEZ, M1-TEZ, IVA, M1-IVA

### Statistical Analyses

#### **Primary Objectives:**

The primary objectives of the study are the evaluation of safety and tolerability, and efficacy of VX-440 in TC with TEZ/IVA (all parts)

The safety endpoints include AEs, clinical laboratory values, 12-lead ECGs, vital signs, and pulse oximetry through the Safety Follow-up Visit (all parts). The safety analysis for all treatment groups in all parts will be descriptive only.

The primary efficacy endpoint is the absolute change from baseline through Day 29 for ppFEV<sub>1</sub> (Parts 1 and 2), 
hypothesis tests will be performed within the mixed-effects model for repeated measures (MMRM) framework at a 5% alpha level, with appropriate adjustment for covariates including stratification factors at randomization. The null within-group hypothesis of no difference in the mean absolute change from baseline through the last on-treatment visit (Day 29 or Week 12) for ppFEV<sub>1</sub>, in all treatment groups, by part, will be tested using a 2-sided 1-sample t test. The adjusted means and 2-sided 95% confidence intervals of the average treatment effects through Day 29 , as applicable, for all within-group and between-group comparisons will be estimated within MMRM.

#### Secondary Objectives:

A secondary objective of the study is the evaluation of the PD effect of VX-440 in TC with TEZ/IVA (all parts)

The PD endpoint is the absolute change in sweat chloride from baseline through Day 29 (Parts 1 and 2)

In Part 1, the null hypothesis of the lack of a decreasing dose-response trend in the mean absolute change from baseline through Day 29 for sweat chloride, between the TC dose groups and placebo will be tested using a multiple comparisons procedure based on the 1-sided maximum *t*-statistic. In all parts, the null within-group hypothesis of no difference in the mean absolute change from baseline through Day 29 for sweat chloride in all treatment groups, by Part, will be

tested using a 2-sided 1-sample *t*-test. The adjusted means and 2-sided 95% confidence intervals of the average treatment effects through Day 29 and between-group comparisons will be estimated within MMRM.

#### Interim Analyses

Separate interim analyses will be performed after:

- all subjects in Part 1 have completed the Safety Follow-up Visit
- all subjects in Part 2 have completed the Safety Follow-up Visit

#### IDMC Reviews

The independent monitoring committee (IDMC) will conduct regular planned safety reviews of study data from all parts of the study as outlined in the IDMC Charter.

### 3 SCHEDULE OF ASSESSMENTS

The schedule of assessments from the Screening Period through the Safety Follow-up Visit are provided in Table 3-1 for Part 1 Cohort 1A, Table 3-2 for Part 1 Cohort 1B, Table 3-3 for Part 2,

All visits will be scheduled relative to the Day 1 Visit (first dose of VX-440 or VX-440 matched placebo).

The CFQ-R assessment must be completed before any other assessment at the clinic visits when it is required. For remaining assessments, assessments may be performed in any order when more than 1 assessment is required at a particular time point. (See Section 11.1.)

Table 3-1 Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1A)

| | Screening | | Treatme | nt Period <sup>b</sup> | | | Safety<br>Follow-up | |
|---|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -28<br>to -1 <sup>d</sup> | Day 1 | Day 8<br>(± 1 day) | Day 15<br>(± 2 days) | Day 29<br>(± 2 days) | Day 43<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | 28 (± 7) Days<br>After Last<br>Dose |
| Informed consent | X | | | | | | | |
| Randomization <sup>e</sup> | | X | | | | | | |
| Demographics | X | | | | | | | |
| Medical history | X | | | | | | | |
| Ophthalmological history | X | | | | | | | |
| CFQ-R <sup>f,g</sup> | | X | | X | X | X | Xh | X |
| Weight <sup>i</sup> | X | X | X | X | X | X | X | X |
| Heighti | X | | | | | | | |
| Vital signs <sup>j</sup> | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>j</sup> | X | X | X | X | X | X | X | X |

All assessments will be performed before dosing, unless noted otherwise. Assessments that are collected before and after dosing will only be collected once if study drug is not administered on the day of the visit (i.e., if subject prematurely discontinued study drug treatment).

- <sup>c</sup> If the subject prematurely discontinues study treatment, an ETT Visit should be scheduled as soon as possible after the decision to terminate study drug treatment. Subjects who prematurely discontinue treatment will also be required to complete the Safety Follow-up Visit. If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit, and a separate Safety Follow-up Visit will not be required.
- All screening results must be reviewed by an appropriately qualified member of the investigator's team before randomization, unless noted otherwise.
- e Randomization may occur on the previous day (Day -1) after all inclusion and exclusion criteria have been confirmed.
- CFQ-R must be completed before the start of any other assessments scheduled at that visit.
- The predose assessment on Day 1 may be performed on the previous day (Day -1) if randomization has occurred.
- b Subjects will complete the CFQ-R at the ETT Visit only if it has been 2 weeks or more since their last visit.
- Weight and height will be measured with shoes off.
- Vital signs and pulse oximetry will be collected after the subject has been seated for at least 5 minutes.

To be eligible to continue into the Treatment Period, subjects must have stable CF disease and have remained on stable CF medication regimen during the 28 days before the Day 1 Visit AND must not have had an acute non-CF illness within 14 days before the Day 1 Visit. See Section 8.1.3.

Table 3-1 Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1A)

| | Screening | | Treatme | nt Period <sup>b</sup> | | | Safety<br>Follow-up | |
|---|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -28<br>to -1 <sup>d</sup> | Day 1 | Day 8<br>(± 1 day) | Day 15<br>(± 2 days) | Day 29<br>(± 2 days) | Day 43<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | 28 (± 7) Days<br>After Last<br>Dose |
| Physical examination <sup>k</sup> | Complete | Abbreviated | | Abbreviated | Abbreviated | | Abbreviated | Complete |
| Ophthalmologic examination <sup>1</sup> | X | | | | | | | |
| Standard 12-lead ECG <sup>m</sup> | X | X | X | X | X | X | X | X |
| Sweat chlorideg,n | X | X | X | X | X | X | X | X |
| Spirometry° | X | X | X | X | X | X | X | X |
| Urinalysisg | X | X | X | X | X | X | X | X |
| Pregnancy test (all females of childbearing potential) | Serum | Urine | | | Urine | | Serum | Serum |
| CFTR genotype <sup>p</sup> | X | | | | | | | |
| FSH <sup>q</sup> | X | | | | | | | |

- Complete and abbreviated PEs are described in Section 11.7.3. Symptom-targeted PEs will occur at any time during the study if triggered by AEs or if deemed necessary by the investigator or healthcare provider.
- The ophthalmological examination can be performed at any time during the Screening Period through the Day 1 Visit (before the first dose of study drug). The screening ophthalmological examination does not have to be performed if there is documentation of an examination that met protocol criteria and was within 3 months before the date of informed consent, or if there is documentation of bilateral lens removal for the subject.
- All standard 12-lead ECGs will be performed after the subject has been seated for at least 5 minutes. On Days 1 and 15, ECGs will be collected before dosing and 4 hours (± 1 hour) after dosing. At all other visits, ECGs will be collected before dosing (as applicable). ECGs collected on Day 1 before dosing will be performed in triplicate.
- Sweat chloride will be measured in all subjects. If the value cannot be determined from the screening test, a sweat chloride value documented in the subject's medical record may be used to establish eligibility.
- Spirometry may be performed pre- or post-bronchodilator at the Screening Visit. Spirometry will be performed pre-bronchodilator, before the morning dose of study drugs, and should be performed at approximately the same time at every other study visit. On Days 1 and 15, spirometry will also be performed pre-bronchodilator 5 hours (± 1 hour) after study drug administration.
- <sup>p</sup> *CFTR* genotyping will be performed for all subjects. If the screening *CFTR* genotype result is not received before randomization, a previous *CFTR* genotype laboratory report may be used to establish eligibility.
- <sup>q</sup> FSH will be measured for any suspected postmenopausal female subjects with at least 12 months of continuous spontaneous amenorrhea.

Table 3-1 Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1A)

| | Screening | | Treatme | nt Period <sup>b</sup> | | | Safety<br>Follow-up | |
|---|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -28<br>to -1 <sup>d</sup> | Day 1 | Day 8<br>(± 1 day) | Day 15<br>(± 2 days) | Day 29<br>(± 2 days) | Day 43<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | 28 (± 7) Days<br>After Last<br>Dose |
| G6PD activity test <sup>r</sup> | X | | | | | | | |
| Serum chemistry and<br>hematology <sup>g</sup> | X | X | X | X | X | X | X | X |
| Coagulationg | X | X | | X | X | | | X |
| PK sampling <sup>t</sup> | | X | X | X | X | X | X | |
| Study drug dosing <sup>u</sup> | | | Day 1 thro | ugh Day 29 | | | | |
| AEs, medications <sup>v</sup> , treatments, and procedures | | | Continuous from | Continuous from signing of the ICF through the Safety Follow-up Visit | | | | |

Blood samples will be collected for PK analysis of VX-440, TEZ, M1-TEZ, IVA, and M1-IVA. On Day 1, samples will be collected before dosing (0 hours) and at 1, 2, 4, and 6 hours after dosing (relative to the morning dose). On Days 8 and 29, a predose sample will be collected before the morning dose of study drug. On Day 15, samples will be collected before dosing (0 hours) and at 1, 2, 4, 6, and 8 hours after dosing. At the Day 43 and the ETT Visits, a single blood sample for PK analysis will be collected.

The last dose of study drug will be the morning dose on Day 29.

v Refer to Section 9.4 for details.

Table 3-2 Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1B)

| | Screening | | Treatment Period | b | | | Safety |
|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -28<br>to -1 <sup>d</sup> | Day 1 | Day 15<br>(± 2 day) | Day 29<br>(± 2 day) | Day 43<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | Follow-up<br>28 (± 7) Days<br>After Last Dose |
| Informed consent | X | | | | | | |
| Randomizatione | | X | | | | | |
| Demographics | X | | | | | | |
| Medical history | X | | | | | | |
| Ophthalmological history | X | | | | | | |
| CFQ-R <sup>f,g</sup> | | X | X | X | X | Xh | X |
| Weight <sup>i</sup> | X | X | X | X | X | X | X |
| Heighti | X | | | | | | |
| Vital signs <sup>j</sup> | X | X | X | X | X | X | X |
| Pulse oximetry <sup>j</sup> | X | X | X | X | X | X | X |

<sup>&</sup>lt;sup>a</sup> All assessments will be performed before dosing, unless noted otherwise. Assessments that are collected before and after dosing will only be collected once if study drug is not administered on the day of the visit (i.e., if subject prematurely discontinued study drug treatment).

- <sup>d</sup> All screening results must be reviewed by an appropriately qualified member of the investigator's team before randomization, unless noted otherwise.
- e Randomization may occur on the previous day (Day -1) after all inclusion and exclusion criteria have been confirmed.
- cFQ-R must be completed before the start of any other assessments scheduled at that visit.
- The predose assessment on Day 1 may be performed on the previous day (Day -1) if randomization has occurred.
- <sup>h</sup> Subjects will complete the CFQ-R at the ETT Visit only if it has been 2 weeks or more since their last visit.
- Weight and height will be measured with shoes off.
- Vital signs and pulse oximetry will be collected after the subject has been seated for at least 5 minutes.

To be eligible to continue into the Treatment Period, subjects must have stable CF disease and have remained on stable CF medication regimen during the 28 days before the Day 1 Visit AND must not have had an acute non-CF illness within 14 days before the Day 1 Visit. See Section 8.1.3.

<sup>&</sup>lt;sup>c</sup> If the subject prematurely discontinues study drug treatment, an ETT Visit should be scheduled as soon as possible after the decision to terminate study drug treatment. Subjects who prematurely discontinue treatment will also be required to complete the Safety Follow-up Visit. If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit, and a separate Safety Follow-up Visit will not be required.

Table 3-2 Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1B)

| | Screening | Treatment Period <sup>b</sup> | | | | | Safety |
|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -28<br>to -1 <sup>d</sup> | Day 1 | Day 15<br>(± 2 day) | Day 29<br>(± 2 day) | Day 43<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | Follow-up<br>28 (± 7) Days<br>After Last Dose |
| Physical examination <sup>k</sup> | Complete | Abbreviated | Abbreviated | Abbreviated | | Abbreviated | Complete |
| Ophthalmologic examination <sup>1</sup> | X | | | | | | |
| Standard 12-lead ECG <sup>m</sup> | X | X | X | X | X | X | X |
| Sweat chloride <sup>g,n</sup> | X | X | X | X | X | X | X |
| Spirometry <sup>o</sup> | X | X | X | X | X | X | X |
| Urinalysis <sup>g</sup> | X | X | X | X | X | X | X |
| Pregnancy test (all females of childbearing potential) | Serum | Urine | | Urine | | Serum | Serum |
| CFTR genotype <sup>p</sup> | X | | | | | | |
| FSH <sup>q</sup> | X | | | | | | |

<sup>&</sup>lt;sup>k</sup> Complete and abbreviated PEs are described in Section 11.7.3. Symptom-targeted PEs will occur at any time during the study if triggered by AEs or if deemed necessary by the investigator or healthcare provider.

The ophthalmological examination can be performed at any time during the Screening Period through the Day 1 Visit (before the first dose of study drug). The screening ophthalmological examination does not have to be performed if there is documentation of an examination that met protocol criteria and was within 3 months before the date of informed consent, or if there is documentation of bilateral lens removal for the subject.

All standard 12-lead ECGs will be performed after the subject has been seated for at least 5 minutes. On Days 1 and 15, ECGs will be collected before dosing and 4 hours (± 1 hour) after dosing. At all other visits, ECGs will be collected before dosing (as applicable). ECGs collected on Day 1 before dosing will be performed in triplicate.

Sweat chloride will be measured in all subjects. If the value cannot be determined from the screening test, a sweat chloride value documented in the subject's medical record may be used to establish eligibility.

Spirometry may be performed pre- or post-bronchodilator at the Screening Visit. Spirometry will be performed pre-bronchodilator, before the morning dose of study drugs, and should be performed at approximately the same time at every other study visit. On Days 1 and 15, spirometry will also be performed pre-bronchodilator, 5 hours (± 1 hour) after study drug administration.

<sup>&</sup>lt;sup>p</sup> *CFTR* genotyping will be performed for all subjects. If the screening *CFTR* genotype result is not received before randomization, a previous *CFTR* genotype laboratory report may be used to establish eligibility.

<sup>&</sup>lt;sup>q</sup> FSH will be measured for any suspected postmenopausal female subjects with at least 12 months of continuous spontaneous amenorrhea.

Table 3-2 Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1B)

| | Screening | | Treatment Period | b | | | Safety |
|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -28<br>to -1 <sup>d</sup> | Day 1 | Day 15<br>(± 2 day) | Day 29<br>(± 2 day) | Day 43<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | Follow-up<br>28 (± 7) Days<br>After Last Dose |
| G6PD activity test <sup>r</sup> | X | | | | | | |
| Serum chemistry and<br>hematology <sup>g</sup> | X | X | X | X | X | X | X |
| Coagulation <sup>g</sup> | X | X | X | X | | | X |
| PK sampling <sup>t</sup> | | X | X | X | X | X | |
| Study drug dosing <sup>u</sup> | | ] | Day 1 through Day 2 | 29 | | | |
| AEs, medications <sup>v</sup> , treatments and procedures | | Conti | nuous from signing ( | of the ICF through | the Safety Follow-u | p Visit | • |

A single blood sample will be collected for the G6PD activity test.

Blood samples will be collected for PK analysis of VX-440, TEZ, M1-TEZ, IVA, and M1-IVA. On Day 1, samples will be collected before dosing (0 hours) and at 1, 2, 4, and 6 hours after dosing (relative to the morning dose). On Day 15, samples will be collected before dosing (0 hours) and at 1, 2, 4, 6, and 8 hours after dosing. On Day 29, a predose sample will be collected before the morning dose of study drug. At the Day 43 and the ETT Visits, a single blood sample for PK analysis will be collected.

<sup>&</sup>lt;sup>u</sup> The last dose of study drug will be the morning dose on Day 29.

v Refer to Section 9.4 for details.

Table 3-3 Study VX15-440-101: Schedule of Assessments for Part 2

| | Screening | Run-in | Period | T | reatment Perio | od <sup>b</sup> | Washou | ıt Period | | Safety<br>Follow, up |
|---|---|---|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -56<br>to -29 <sup>e</sup> | Day -28<br>(± 1 day) | Day -14 <sup>f</sup><br>(± 1 day) | Day 1 | Day 15<br>(± 2 days) | Day 29<br>(± 2 days) | Day 43 (± 3 days) | Day 57<br>(± 3 days) | ETT<br>Visit <sup>e</sup> | Follow-up<br>28 (± 7) Days<br>After Last<br>Dose <sup>d</sup> |
| Informed consent | X | | | | | | | | | |
| Randomization <sup>g</sup> | | | | X | | | | | | |
| Demographics | X | | | | | | | | | |
| Medical history | X | | | | | | | | | |
| Ophthalmological<br>history | X | | | | | | | | | |
| CFQ-R <sup>h,i</sup> | | | | X | X | X | X | X | $X^{j}$ | X |
| Weight <sup>k</sup> | X | X | | X | X | X | X | X | X | X |
| Height <sup>k</sup> | X | | | | | | | | | |
| Vital signs <sup>1</sup> | X | X | | X | X | X | X | X | X | X |
| Pulse oximetry <sup>1</sup> | X | X | | X | X | X | X | X | X | X |

- All assessments will be performed before dosing, unless noted otherwise. Assessments that are collected before and after dosing will only be collected once if study drug is not administered on the day of the visit (i.e., if subject prematurely discontinued study drug treatment).
- To be eligible to continue into the Treatment Period, subjects must have stable CF disease and have remained on stable CF medication regimen during the 28 days before the Day 1 Visit AND must not have had an acute non-CF illness within 14 days before the Day 1 Visit. See Section 8.1.3.
- <sup>c</sup> If the subject prematurely discontinues study treatment, an ETT Visit should be scheduled as soon as possible after the decision to terminate study drug treatment. Subjects who prematurely discontinue treatment will also be required to complete the Safety Follow-up Visit. If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit, and a separate Safety Follow-up Visit will not be required.
- <sup>d</sup> Part 2 subjects who meet criteria specified in Section 8.1.5 will not have a Safety Follow-up Visit.
- <sup>e</sup> All screening results must be reviewed by an appropriately qualified member of the investigator's team before the subject receives the first dose of TEZ/IVA in the Run-in Period on Day -28, unless noted otherwise.
- The Day -14 Visit is only required for subjects who are naïve to TEZ/IVA treatment.
- Randomization may occur on the previous day (Day -1) after all inclusion and exclusion criteria and criteria for entry into the Treatment Period have been confirmed. See Section 8.1.3.
- <sup>h</sup> CFQ-R must be completed before the start of any other assessments scheduled at that visit.
- The predose assessment on Day 1 may be performed on the previous day (Day -1) if randomization has occurred.
- Subjects will complete the CFQ-R at the ETT Visit only if it has been 2 weeks or more since their last visit.
- Weight and height will be measured with shoes off.
- Vital signs and pulse oximetry will be collected after the subject has been seated for at least 5 minutes.

Table 3-3 Study VX15-440-101: Schedule of Assessments for Part 2

| | Screening | Run-in | Period | Tr | eatment Perio | od <sup>b</sup> | Washou | t Period | | Safety<br>Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -56<br>to -29 <sup>e</sup> | Day -28<br>(± 1 day) | Day -14 <sup>f</sup><br>(± 1 day) | Day 1 | Day 15<br>(± 2 days) | Day 29<br>(± 2 days) | Day 43<br>(± 3 days) | Day 57<br>(± 3 days) | ETT<br>Visit° | 28 (± 7) Days<br>After Last<br>Dose <sup>d</sup> |
| Physical<br>examination <sup>m</sup> | Complete | Abbreviated | | Abbreviated | Abbreviated | Abbreviated | | Abbreviated | Abbreviated | Complete |
| Ophthalmologic<br>examination <sup>n</sup> | X | | | | | | | | | |
| Standard 12-lead<br>ECG° | X | X | | X | X | X | X | X | X | X |
| Sweat chloride <sup>i,p</sup> | X | | X | X | X | X | X | X | X | |
| Spirometry <sup>q</sup> | X | | X | X | X | X | X | X | X | X |
| Urinalysis <sup>i</sup> | X | X | | X | X | X | X | X | X | X |
| Pregnancy test (all<br>females of<br>childbearing<br>potential) | Serum | Urine | | Urine | | Urine | | Urine | Serum | Serum |
| CFTR genotype <sup>r</sup> | X | | | | | | | | | |
| FSH <sup>s</sup> | X | | | | | | | | | |

- Complete and abbreviated PEs are described in Section 11.7.3. Symptom-targeted PEs will occur at any time during the study if triggered by AEs or if deemed necessary by the investigator or healthcare provider.
- The ophthalmological examination can be performed at any time during the Screening Period through the Day 1 Visit (before the first dose of study drug). The screening ophthalmological examination does not have to be performed if there is documentation of an examination that met protocol criteria and was within 3 months before the date of informed consent, or if there is documentation of bilateral lens removal for the subject.
- All standard 12-lead ECGs will be performed after the subject has been seated for at least 5 minutes. On Days 1 and 15, ECGs will be collected before dosing and 4 hours (± 1 hour) after dosing. At all other visits, ECGs will be collected before dosing (as applicable). ECGs collected on Day 1 before dosing will be performed in triplicate.
- Sweat chloride will be measured in all subjects. If the value cannot be determined from the screening test, a sweat chloride value documented in the subject's medical record may be used to establish eligibility.
- Spirometry may be performed pre- or post-bronchodilator at the Screening Visit. Spirometry will be performed pre-bronchodilator, before the morning dose of study drugs, and should be performed at approximately the same time at every other study visit. On Days 1 and 15, spirometry will also be performed pre-bronchodilator, 5 hours (± 1 hour) after study drug administration.
- <sup>r</sup> *CFTR* genotyping will be performed for all subjects. If the screening *CFTR* genotype result is not received before Day -28, a previous *CFTR* genotype laboratory report may be used to establish eligibility.

Table 3-3 Study VX15-440-101: Schedule of Assessments for Part 2

| | Screening | Run-in | Period | Tı | eatment Perio | od <sup>b</sup> | Washou | t Period | | Safety<br>Follow, up |
|---|---|---|---|---|---|---|---|---|---|---|
| Event/Assessment <sup>a</sup> | Days -56<br>to -29° | Day -28<br>(± 1 day) | Day -14 <sup>f</sup><br>(± 1 day) | Day 1 | Day 15<br>(± 2 days) | Day 29<br>(± 2 days) | Day 43<br>(± 3 days) | Day 57<br>(± 3 days) | ETT<br>Visit <sup>c</sup> | Follow-up<br>28 (± 7) Days<br>After Last<br>Dose <sup>d</sup> |
| G6PD activity test <sup>t</sup> | X | | | | | | | | | |
| Serum chemistry<br>and hematology <sup>i</sup> | X | X | | X | X | X | X | X | X | X |
| Coagulation <sup>i</sup> | X | X | | X | X | X | | | | X |
| PK sampling <sup>v</sup> | | | | X | X | X | X | | X | |
| TEZ/IVA dosing <sup>w</sup> | | | | Day | -28 through D | ay 57 | | | | |
| VX-440 or placebo<br>dosing <sup>x</sup> | | | | Day | / 1 through Da | y 29 | | | | |
| AEs, medications <sup>y</sup> ,<br>treatments and<br>procedures | | Continuous from signing of the ICF through the Safety Follow-up Visit | | | | | | | | |

FSH will be measured for any suspected postmenopausal female subjects with at least 12 months of continuous spontaneous amenorrhea.

t A single blood sample will be collected for the G6PD activity test

Blood samples will be collected for PK analysis of VX-440, TEZ, M1-TEZ, IVA, and M1-IVA. On Day 1, samples will be collected before dosing (0 hours) and at 1, 2, 4, and 6 hours after dosing (relative to morning dose). On Day 15, samples will be collected before dosing (0 hours) and at 1, 2, 4, 6, and 8 hours after dosing. On Day 29, a predose sample will be collected before the morning dose of study drug. At the Day 43 Visit, a single blood sample for PK analysis will be collected before the morning dose of TEZ/IVA. At the ETT Visit, a single blood sample for PK analysis will be collected.

The last dose of TEZ/ivacaftor will be the morning dose on Day 57.

The last dose of VX-440 or placebo will be the morning dose on Day 29.

y Refer to Section 9.4 for details.

## 4 TABLE OF CONTENTS

| 1 | Title Page | 1 |
|----|--------------------------------------------------------|------|
| 2 | Protocol Synopsis | |
| 3 | Schedule of Assessments | . 10 |
| 4 | Table of Contents | |
| | List of Tables. | |
| | List of Figures | |
| | Glossary of Terms | |
| 5 | Introduction | |
| | 5.1 Background | |
| | 5.2 Rationale for the Present Study | |
| 6 | Study Objectives | |
| | 6.1 Primary Objectives | |
| _ | 6.2 Secondary Objectives | |
| 7 | Study Endpoints | |
| | 7.1 Primary Endpoints | |
| | 7.2 Secondary Endpoints | . 32 |
| 8 | Study Design | 32 |
| 0 | 8.1 Overview of Study Design | |
| | 8.1.1 Screening | |
| | 8.1.1.1 Repetition of Screening Assessment(s) | |
| | 8.1.1.2 Rescreening | |
| | 8.1.1.3 Extension of Screening Period Window | |
| | 8.1.2 Run-in Period (Part 2) | |
| | 8.1.3 Treatment Period | |
| | 8.1.4 Washout Period (Part 2) | |
| | 8.1.5 Follow-up | . 38 |
| | 8.1.6 Early Termination of Treatment | . 39 |
| | 8.1.7 Independent Data Monitoring Committee | . 39 |
| | 8.2 Rationale for Study Design and Study Drug Regimens | |
| | 8.2.1 Study Design | |
| | 8.2.2 Study Drug Dose and Duration | |
| | 8.2.3 Rationale for Study Population. | |
| | 8.2.4 Rationale for Study Assessments | |
| 9 | Study Population | |
| | 9.1 Inclusion Criteria | |
| | 9.2 Exclusion Criteria | |
| | 9.3 Prohibited Medications | |
| | 9.4 Prior and Concomitant Medications | |
| | 9.5 Removal of Subjects | |
| 10 | 9.6 Replacement of Subjects | |
| 10 | Study Drug Administration and Management | |
| | 10.1 Preparation and Dispensing | . 48 |

| | 10.2 Adr | ninistration | 48 |
|----|-----------|----------------------------------------------------|----|
| | 10.2.1 | Missed Doses | 49 |
| | 10.3 Met | thod of Assigning Subjects to Treatment Groups | 49 |
| | | dy Drug Interruption and Stopping Rules | |
| | | kaging and Labeling | |
| | | dy Drug Supply, Storage, and Handling | |
| | | g Accountability | |
| | | posal, Return, or Retention of Unused Drug | |
| | | npliance | |
| | | nding and Unblinding | |
| | | Blinding | |
| | | Unblinding | |
| 11 | | ients | |
| | | ning of Assessments | |
| | 11.2 Sub | ect and Disease Characteristics | 54 |
| | 11.3 Pha | rmacokinetics | 54 |
| | 11.3.1 | Blood Sampling | |
| | 11.3.2 | Processing and Handling of Pharmacokinetic Samples | 55 |
| | 11.3.3 | Bioanalysis | |
| | | rmacodynamics | |
| | 11.4.1 | Sweat Chloride | 55 |
| | 11.6 Effi | cacy | 55 |
| | 11.6.1 | Spirometry | 55 |
| | 11.6.2 | Height and Weight | |
| | 11.6.3 | Cystic Fibrosis Questionnaire-Revised | 57 |
| | 11.7 Safe | ety | 58 |
| | 11.7.1 | Adverse Events | 58 |
| | 11.7.2 | Clinical Laboratory Assessments | 58 |
| | 11.7.3 | Physical Examinations and Vital Signs | 60 |
| | 11.7.4 | Pulse Oximetry | 60 |
| | 11.7.5 | Electrocardiograms | 60 |
| | 11.7.6 | Ophthalmologic Examination | 61 |
| | 11.7.7 | Contraception and Pregnancy | 61 |
| | 11.7. | 7.1 Contraception | 62 |
| | 11.7. | 7.2 Pregnancy | 63 |
| 12 | Statistic | cal and Analytical Plans | 63 |
| | 12.1 San | aple Size and Power | 63 |
| | 12.1.1 | Primary Objectives | 63 |
| | 12.1. | 1.1 Safety and Tolerability | 63 |
| | 12.1. | 1.2 Efficacy | 64 |
| | 12 1 2 | Secondary Objectives | 6/ |

| 12.1.2.1 | Pharmacodynamic Effect (Part 1) | 64 |
|---|---|---|
| 12.2 Analysis | s Sets | 66 |
| | al Analysis | |
| 12.3.1 Ge | neral Considerations | 66 |
| 12.3.2 Bac | ckground Characteristics | 67 |
| 12.3.2.1 | | 67 |
| 12.3.2.2 | Demographics and Baseline Characteristics | 67 |
| 12.3.2.3 | Prior and Concomitant Medications | |
| 12.3.2.4 | Study Drug Exposure and Compliance | |
| 12.3.2.5 | Important Protocol Deviations | 68 |
| 12.3.3 Eff | icacy Analysis | 68 |
| 12.3.3.1 | Analysis of Primary Efficacy Variables | 68 |
| 12.3.3.2 | Analysis of Secondary Efficacy Variables | |
| 12.3.4 Pha | armacodynamic Analysis | 69 |
| | Pharmacodynamic Effect | |
| 12.3.5 Saf | fety Analysis | 70 |
| 12.3.5.1 | Adverse Events | 70 |
| 12.3.5.2 | Clinical Laboratory Assessments | 71 |
| 12.3.5.3 | Electrocardiogram | 71 |
| 12.3.5.4 | Vital Signs | 71 |
| 12.3.5.5 | Pulse Oximetry | 72 |
| 12.3.5.6 | Physical Examination. | 72 |
| 12.3.5.7 | Other Safety Analysis | 72 |
| 12.3.6 Into | erim and IDMC Analyses | 72 |
| 12.3.6.1 | Interim Analysis | 72 |
| 12.3.6.2 | IDMC Analysis | 72 |
| 12.4 Clinical | Pharmacology Analysis | 72 |
| 12.4.1 Pha | armacokinetic Analysis | 72 |
| 12.4.2 Pha | armacokinetic/Pharmacodynamic Analyses | 72 |
| 13 Procedural, | Ethical, Regulatory, and Administrative Considerations | 73 |
| | Event and Serious Adverse Event Documentation, Severity Grading, and | |
| Reportii | ng | 73 |
| | verse Events | |
| 13.1.1.1 | Definition of an Adverse Event. | 73 |
| 13.1.1.2 | Clinically Significant Assessments | 73 |
| 13.1.1.3 | Documentation of Adverse Events | 73 |
| 13.1.1.4 | Adverse Event Severity | 74 |
| 13.1.1.5 | Adverse Event Causality | 75 |
| 13.1.1.6 | Study Drug Action Taken | 75 |
| 13.1.1.7 | Adverse Event Outcome | |
| 13.1.1.8 | Treatment Given | 76 |
| 13.1.2 Ser | rious Adverse Events | |
| 13.1.2.1 | Definition of a Serious Adverse Event | |
| 13.1.2.2 | Documentation of Serious Adverse Events | 77 |
| 13 1 2 3 | Reporting Serious Adverse Events | 77 |

| 13.1.2.4 Expedited Reporting and Investigator Safety Letters | 77 |
|---|---|
| 13.2 Administrative Requirements | 77 |
| 13.2.1 Ethical Considerations | 77 |
| 13.2.2 Subject Information and Informed Consent | 78 |
| 13.2.3 Investigator Compliance | |
| 13.2.4 Access to Records | |
| 13.2.5 Subject Privacy | |
| 13.2.6 Record Retention | |
| 13.2.7 Study Termination | |
| 13.3 Data Quality Assurance | |
| 13.4 Monitoring | |
| 13.5 Electronic Data Capture | |
| 13.6 Publications and Clinical Study Report | |
| 13.6.2 Clinical Study Report | 81 |
| 14 References | |
| APPENDIX A <i>CFTR</i> Mutations That Are Predicted to Result in a CFTR Pr | |
| Minimal Function (Part 1 | |
| 15 Protocol Signature Pages | 87 |
| 15.1 Sponsor Signature Page | |
| 15.2. Investigator Signature Page | 88 |

### **List of Tables**

| Table 3-1 | Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1A) | 11 |
|---|---|---|
| Table 3-2 | Study VX15-440-101: Schedule of Assessments for Part 1 (Cohort 1B) | |
| Table 3-3 | Study VX15-440-101: Schedule of Assessments for Part 2 | 17 |
| Table 8-1 | Key Study Elements by Part | |
| Table 8-2 | Treatment Arms and Planned Doses by Part | 34 |
| Table 9-1 | Prohibited Medications | 46 |
| Table 10-1 | Study Drug | |
| Table 11-1 | Acceptable Pharmacokinetic Sampling Windows | 54 |
| Table 11-2 | Safety Laboratory Test Panels | 59 |
| Table 11-3 | Contraceptive Requirements | 62 |
| Table 12-1 | Probability of Observing an Adverse Event | 63 |
| Table 12-2 | Power for Within-group Difference for Mean Absolute Change From Base | |
| | ppFEV <sub>1</sub><br>Contrast Coefficients for the Multiple Comparisons Procedure in Part 1, C | 64 |
| Table 12-3 | Contrast Coefficients for the Multiple Comparisons Procedure in Part 1, C | ohort |
| | 1B | |
| Table 12-4 | Power to Detect a Dose-response Trend Based on Change From Baseline | in Sweat |
| | Chloride in Part 1, Cohort 1B | 65 |
| Table 12-5 | Power for Within-group Difference for Mean Absolute Change From Base | eline in |
| | Sweat Chloride | |
| Table 13-1 | Grading of AE Severity | 74 |
| Table 13-2 | Classifications for AE Causality | 75 |
| Table 13-3 | Classifications for Study Drug Action Taken With Regard to an AE | 75 |
| Table 13-4 | Classifications for Outcome of an AE | 75 |
| List of Figu | ures | |
| Figure 8-1 | Schematic of the Study Design for Parts 1 and 2 | 35 |

# **Glossary of Terms**

| Olossary or re | |
|---|---|
| Abbreviation | Term |
| AE | adverse event |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransaminase |
| BMI | body mass index |
| CF | cystic fibrosis |
| CFQ-R | Cystic Fibrosis Questionnaire-Revised |
| CFTR | CF transmembrane conductance regulator protein |
| CPAP | clinical pharmacology analysis plan |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTFG | Clinical Trial Facilitation Group |
| CYP | cytochrome P450 |
| ECG | electrocardiogram |
| EDC | electronic data capture |
| ETT | early termination of treatment |
| F508del | CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein (make italics) |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FEV <sub>1</sub> | forced expiratory volume in 1 second |
| FSH | follicle-stimulating hormone |
| G6PD | glucose-6-phosphate dehydrogenase |
| GCP | Good Clinical Practice |
| GPS | Global Patient Safety |
| HBE | human bronchial epithelial |
| HMA | Heads of Medicines Agencies |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IDMC | independent data monitoring committee |
| IEC | independent ethics committee |
| INN | international nonproprietary name |
| IPD | important protocol deviation |
| IRB | institutional review board |
| IVA | ivacaftor |
| IWRS | interactive web response system |
| LFT | liver function test |
| LUM | lumacaftor |
| max | maximum value |

| Abbreviation | Term |
|--------------|--------------------------------------------------------|
| MBW | multiple-breath washout |
| MCP | multiple comparisons procedure |
| MF | minimum function |
| min | minimum value |
| MMRM | mixed-effects model for repeated measures |
| N | total sample size (e.g., number of subjects treated) |
| NA | not applicable |
| OATP1B1 | organic anion transporting polypeptide 1B1 |
| OATP1B3 | organic anion transporting polypeptide 1B3 |
| P | probability |
| PD | pharmacodynamic, pharmacodynamics |
| PE | physical examination |
| PK | pharmacokinetic, pharmacokinetics |
| $ppFEV_1$ | percent predicted forced expiratory volume in 1 second |
| q12h | every 12 hours |
| qd | daily |
| QTc | QT interval corrected |
| QTcF | QT interval corrected by Fridericia's formula |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SE | standard error |
| TBD | to be determined |
| TC | triple combination |
| TE | treatment-emergent |
| TEAE | treatment-emergent adverse event |
| TEZ | tezacaftor |
| ULN | upper limit of normal |
| USAN | United States adopted name |
| Vertex | Vertex Pharmaceuticals Incorporated |

#### 5 INTRODUCTION

### 5.1 Background

Cystic fibrosis (CF) affects more than 70,000 children and adults worldwide<sup>1</sup> and is the most common fatal genetic disease in persons of European descent.<sup>2</sup> Based on its prevalence, CF qualifies as an orphan disease.<sup>3,4</sup> CF is caused by a defect in the gene encoding the CF transmembrane conductance regulator (CFTR), an ion channel that regulates the flow of chloride and other ions in epithelia of various tissues, including lungs, pancreas and other gastrointestinal organs, and sweat glands.<sup>2</sup> Decreased CFTR activity in people with CF results in multisystem pathology<sup>5</sup>, beginning at birth. Despite progress in the treatment of CF with antibiotics and mucolytics, the median predicted survival age for a person with CF is approximately 40 years.<sup>2,6</sup> More effective treatments are needed for CF.

To address this medical need, Vertex Pharmaceuticals Incorporated is developing treatment regimens that include CFTR modulators to target the underlying cause of CF: the defective CFTR protein. Two types of CFTR modulators have been developed: potentiators, which increase the channel gating activity of the CFTR protein, and correctors, which increase the quantity of CFTR at the cell surface. Because potentiators can increase the activity of CFTR protein delivered to the cell surface by correctors, CFTR potentiators and correctors are complementary therapeutic approaches.

Ivacaftor (IVA; Kalydeco®), the first CFTR modulator developed by Vertex, is an orally administered CFTR potentiator that increases the channel-open probability of CFTR protein to enhance chloride transport. Globally, Kalydeco is indicated for the treatment of CF in patients as young as 2 years who have the *G551D* and certain other gating mutations, as well as the *R117H* mutation in the *CFTR* gene in certain regions.<sup>7</sup>

Lumacaftor (LUM; VX-809) and tezacaftor (TEZ; VX-661) are orally administered first-generation CFTR correctors developed by Vertex that act directly on CFTR to improve its cellular processing and trafficking, thereby increasing the quantity of functional F508del-CFTR protein at the cell surface. *F508del*, the most prevalent mutation in people with CF, occurs in about 83% of CF patients of European descent, and results in a decreased quantity of CFTR protein at the cell surface. Orkambi™ (LUM/IVA combination therapy) is approved in the US, EU, Canada, and Australia for patients 12 years and older who are homozygous for *F508del*. Phase 3 studies of TEZ/IVA combination therapy are ongoing in populations that are homozygous or heterozygous for *F508del*.

VX-440 is a second-generation CFTR corrector that acts through a different site of the CFTR protein than LUM and TEZ. In vitro, VX-440 improves the processing and trafficking of F508del-CFTR, thereby increasing the quantity of functional F508del-CFTR protein at the cell surface. VX-440 has been studied in vitro in combination with the first generation corrector TEZ. Consistent with different mechanisms of action, the effects of VX-440 and TEZ are additive. The activity of the CFTR protein delivered to the cell surface by VX-440, alone or in combination with TEZ, is potentiated by IVA. In human bronchial epithelial (HBE) cells derived from CF patients homozygous for *F508del*, the triple combination (TC) of VX-440, TEZ, and IVA increased CFTR-mediated chloride transport more than the dual combinations (VX-440 and TEZ; VX-440 and IVA; TEZ and IVA) or individual agents (VX-440; TEZ; IVA). These data, as

well as the nonclinical pharmacokinetic (PK) and safety profile, support the development of VX-440 in combination with other CFTR modulators for the treatment of CF.

### 5.2 Rationale for the Present Study

The present study is the first clinical study of VX-440 in subjects with CF and is designed to evaluate the safety and efficacy of VX-440 in triple combination with TEZ and IVA.

VX-440 has been studied in vitro and in vivo, and the safety profile in the nonclinical toxicology studies supports continued development of VX-440 with appropriate measures given the potential for teratogenicity.<sup>8,9</sup>

The safety, tolerability, and PK of VX-440 as monotherapy or in TC with TEZ/IVA are being evaluated in healthy subjects (Study VX15-440-001 [Study 001] and VX16-440-002 [Study 002]). Single doses of VX-440 up to 1600 mg and multiple doses of VX-440 up to 600 mg q12h have been generally safe and well tolerated. Multiple doses of VX-440 up to 600 mg q12h in TC with TEZ (100 mg qd) and IVA (up to 300 mg q12h) were also safe and well tolerated.

Based on the data from nonclinical and clinical studies of VX-440, TEZ, and IVA to date and the current unmet medical need for new treatments for CF, there is potential for benefit to CF patients from the development of this treatment. Therefore, the overall risk-benefit balance for this study is considered to be acceptable.

#### 6 STUDY OBJECTIVES

### 6.1 Primary Objectives

- To evaluate the safety and tolerability of VX-440 in and IVA
- To evaluate the efficacy of VX-440 in triple combination with TEZ and IVA

## 6.2 Secondary Objectives

- To evaluate the pharmacodynamic (PD) effect of VX-440 in TEZ and IVA on sweat chloride concentrations
- To evaluate the PK of VX-440 when administered in and IVA
- To evaluate the PK of TEZ, IVA, and their respective metabolites when administered with VX-440

#### 7 STUDY ENDPOINTS

## 7.1 Primary Endpoints

- Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values, standard 12-lead electrocardiograms (ECGs), vital signs, and pulse oximetry
- Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline through Day 29 (Parts 1 and 2)

## 7.2 Secondary Endpoints

| Absolute change in sweat chloride concentration 2) | s from baseline through Day 29 (Parts 1 and |
|---|---|
| <ul> <li>Relative change in ppFEV<sub>1</sub> from baseline through</li> </ul> | h Day 29 (Parts 1 and 2) |
| PK parameters of VX-440, TEZ, M1-TEZ, IVA | and M1-IVA |
| 8 STUDY DESIGN | |
| 8.1 Overview of Study Design | |
| This is a Phase 2, randomized, double-blind, placebound multicenter study designed to evaluate the safety and combination with TEZ and IVA. | |
| Approximately 198 subjects with CF will be enrolle Parts 1 will be sequential, while enrollment of 1B. | d across Parts 1 . Enrollment of Part 2 will be in parallel with Part 1 Cohort |
| Part 1 will consist of 2 cohorts: Cohort 1A and Cohort 1B will be sequential. After all Cohort 1A sureview of all available safety and PK data will be coinvestigator(s). Dosing of Cohort 1B will begin after and PK data. | bjects complete the Day 15 Visit, a blinded nducted by the Vertex study team and lead |
| Part 2 will initiate after the Cohort 1A blinded revie | ew, if supported by safety and PK data. |

Key study elements of each part are summarized in Table 8-1. The treatment arms and randomization ratios for each part are summarized in Table 8-2. A schematic of the study design is shown in Figure 8-1 (Parts 1 and 2)

Interim analyses are described in Section 12.3.6.1.

All parts of this study will include a Screening Period, Treatment Period, and Safety Follow-up Visit. Part 2 will also include a 4-week Run-in Period and a 4-week Washout Period after the Treatment Period.

Table 8-1 Key Study Elements by Part

| | <u> </u> | |
|---|---|---|
| | Part 1 <sup>a</sup> | Part 2 |
| Genotype | F508del/MF | F508del/F508del |
| Age | ≥18 years | ≥18 years |
| ppFEV <sub>1</sub> criteria | ≥40 to ≤90 | ≥40 to ≤90 |
| Number of subjects | s Approximately 42 <sup>a</sup> | Approximately 24 |
| Stratification c | ppFEV <sub>1</sub> <sup>d</sup> | $ppFEV_1$ |
| | • ≥70 | • ≥70 |
| | • <70 | • <70 |
| Study design | Parallel | Parallel |
| Comparator | Placebo | TEZ/IVA |
| VX-440 treatment | 4 weeks | 4 weeks |
| duration | | |

IVA: ivacaftor; MF: minimal function; ppFEV<sub>1</sub>: percent predicted forced expiratory volume in 1 second; q12h: every 12 hours; TC: triple combination; TEZ: tezacaftor

- Additional stratification information is provided in Section 8.1.3.
- Stratification will be conducted for Cohort 1B subjects only.

Part 1 consists of Cohort 1A and Cohort 1B. Approximately 10 subjects will be in Cohort 1A and approximately 32 subjects will be in Cohort 1B

Table 8-2 Treatment Arms and Planned Doses by Part

| Part | | | TEZ | IVA |
|---|---|---|---|---|
| Randomization ratio | Treatment Arm | VX-440 Dosage | Dosage | Dosage |
| Part 1 Cohort 1A | TC-1A | 200 mg q12h | 100 mg qd | 150 mg q12h |
| 4:1 | Triple placebo | Placebo | Placebo | Placebo |
| Part 1 Cohort 1B | TC-1B-high | 600 mg q12h <sup>a</sup> | 50 mg q12h | 300 mg q12h <sup>a</sup> |
| 2:1:1 | TC-1B-low | 200 mg q12h | 50 mg q12h | 150 mg q12h |
| | Triple placebo | Placebo | Placebo | Placebo |
| Part 2 <sup>b</sup> | TC-2 | 600 mg q12h <sup>a</sup> | 50 mg q12h | 300 mg q12h <sup>a</sup> |
| 3:1 | TEZ/IVA | Placebo | 100 mg qd | 150 mg q12h |

In the "TC-1B-high" and "TC-2" treatment arms, the dosage of VX-440 will be determined based on safety and PK data from Cohort 1A. The planned dose is shown, but may be reduced to 400 mg q12h.

In Part 2, all subjects will also receive TEZ 100 mg qd/IVA 150 mg q12h during the Run-in Period and the Washout Period.

Figure 8-1 Schematic of the Study Design for Parts 1 and 2

**Part 1 Cohort 1A:** *F508del*/MF (N ~ 10)

Randomization: 4:1



Part 1 Cohort 1B: F508del/MF (N ~ 32)

Randomization: 2:1:1

Stratification: ppFEV<sub>1</sub>:  $\geq$ 70 versus <70



Part 2: F508del/F508del (N ~ 24)

Randomization: 3:1

Stratification: ppFEV<sub>1</sub>:  $\geq$ 70 versus <70



IVA: ivacaftor; MF: minimal function; N: number of subjects; ppFEV<sub>1</sub>: percent predicted forced expiratory volume in 1 second; q12h: every 12 hours; qd: daily; TEZ: tezacaftor; TC: triple combination

Notes: Schematic is not drawn to scale. TC includes VX-440, TEZ, and IVA. The dose of each component of the TC is shown by treatment arm in Table 8-2. In Part 2, the dose of TEZ/IVA during the Run-in Period and the Washout Period will be TEZ 100 mg qd/IVA 150 mg q12h. Additional stratification information is provided in Section 8.1.3.



Study visits and assessments to be conducted are shown in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2),

### 8.1.1 Screening

For Parts 1 the Screening Period will occur within 28 days before the first dose of study drug in the Treatment Period. For Part 2, the Screening Period will occur within 28 days before the first dose of TEZ/IVA in the Run-in Period.

Assessments to be conducted will be used to confirm that subjects meet the eligibility criteria for the study. The investigator (or an appropriate authorized designee) will obtain informed consent and assent, if applicable, from each subject before any study procedure takes place.

The screening ophthalmologic examination does not have to be performed if there is documentation of an examination that met protocol criteria and was within 3 months before the date of informed consent (or assent, when applicable; Section 11.7.6) or if there is documentation of bilateral lens removal for the subject.
# 8.1.1.1 Repetition of Screening Assessment(s)

Repetition of individual screening assessment(s) that did not meet eligibility criteria is not permitted with the following exceptions:

- If there is clear evidence of a laboratory error (e.g., hemolyzed sample) or equipment malfunction, collection of a repeat sample for the appropriate laboratory test or assessment may be permitted with the approval of the medical monitor.
- Exclusionary liver function test (LFT) levels, which may be retested once within 14 days of the original screening date, with approval of the medical monitor.

If screening spirometry measurements fail to meet acceptability and repeatability criteria as specified by American Thoracic Society/European Respiratory Society guidelines<sup>10</sup>, repeat spirometry evaluation may be performed once.

If repeat values of the individual assessment(s) are within the eligibility criteria and completed within the screening window, then the subject is eligible for the study.

### 8.1.1.2 Rescreening

Subjects may only be rescreened with the approval of the medical monitor. If a subject is rescreened, all screening assessments will be repeated except for *CFTR* genotyping, follicle-stimulating hormone (FSH) level (if serum FSH level was ≥40 mIU/mL during prior screening), G6PD activity test (if total bilirubin level was <2 × upper limit of normal [ULN] during prior screening), sweat chloride level, and the ophthalmologic examination (if documentation shows it was performed within the last 3 months). If a subject is rescreened, the new screening window will begin once the first rescreening assessment has been initiated.

## 8.1.1.3 Extension of Screening Period Window

A subject may have the Screening Period window extended by 2 weeks, without medical monitor approval, for the following reasons:

- Repetition of the Screening Period assessments (Section 8.1.1.1)
- Unexpected operational or logistic delays, or to meet the eligibility criteria
- Scheduling of ophthalmologic examination (Section 11.7.6)
- Repetition of spirometry assessment if results are of poor quality

A subject may have the Screening Period window extended by 4 weeks, without medical monitor approval, for the following reason:

• For Parts 1 subjects, washout of TEZ/IVA during the Screening Period if enrolling from Study VX14-661-110 (Study 661-110)

### 8.1.2 Run-in Period (Part 2)

The Run-in Period will have a total duration of 4 weeks and is designed to establish a reliable ontreatment (TEZ/IVA) baseline for the Treatment Period. Subjects will receive TEZ 100 mg qd/IVA 150 mg q12h during the Run-in Period. The first dose of TEZ/IVA will be administered at the Day -28 Visit. The last dose of TEZ/IVA within the Run-in Period will be administered on Day -1 (1 day before the Day 1 Visit).

### 8.1.3 Treatment Period

The Treatment Period will last approximately 4 weeks for Parts 1 and 2, Study drug administration details are provided in Section 10.2.

For all parts, subjects must meet both of the following criteria to continue into the Treatment Period:

- Must have stable CF disease (as judged by the investigator) and have remained on a stable CF medication regimen during the 28 days before the Day 1 Visit. (For example, subjects cannot have an acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy [including antibiotics] for pulmonary disease within 28 days before the Day 1 Visit.)
- Must not have had an acute non-CF illness (e.g., gastroenteritis) within the 14 days before the Day 1 Visit.

If these criteria are not met, subjects may not be randomized and enter into the Treatment Period.

Randomization will occur before the first dose of study drug during the Treatment Period and may occur on Day 1 or Day -1 after all inclusion and exclusion criteria and the criteria for entry into the Treatment Period have been confirmed. Randomization will be stratified according to the criteria shown in Table 8-1. For ppFEV<sub>1</sub> stratification, Day -14 values will be used for subjects in Part 2 who are naïve to TEZ/IVA treatment, while screening ppFEV<sub>1</sub> values will be used for all other subjects, including subjects in Parts 1

For Part 2, subjects who prematurely discontinue TEZ/IVA during the Run-in Period will not be randomized or participate in the Treatment Period.



# 8.1.4 Washout Period (Part 2)

The Washout Period will last approximately 4 weeks and is designed to allow for the measurement of VX-440 off-treatment effects. Subjects will receive TEZ 100 mg qd/IVA 150 mg q12h during the Washout Period.

#### 8.1.5 Follow-up

There will be an outpatient Safety Follow-up Visit occurring approximately 28 days after the last dose of study drug for subjects who complete study drug dosing and for subjects who prematurely discontinue study drug dosing.

The following Part 2 subjects will not have a Safety Follow-up Visit:

- Part 2 subjects who do not meet the criteria to enter the Treatment Period (Section 8.1.3), and re-enter Study 661-110
- Part 2 subjects who complete the Day 57 Visit and re-enter Study 661-110

All other Part 2 subjects will have a Safety Follow-up Visit.

### 8.1.6 Early Termination of Treatment

If a subject prematurely discontinues treatment, an Early Termination of Treatment (ETT) Visit should be scheduled as soon as possible after the decision to terminate study drug treatment. Subjects who prematurely discontinue treatment will also be required to complete the Safety Follow-up Visit, approximately 28 days after their last dose of study drug.

If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit, and a separate Safety Follow-up Visit will not be required.



If a subject withdraws from the study and also withdraws consent for disclosure of future information, no further evaluations should be performed and no additional data should be collected. Vertex may retain and continue to use any data collected before such withdrawal of consent.

# 8.1.7 Independent Data Monitoring Committee

This study will be monitored by an external independent data monitoring committee (IDMC), which will conduct periodic reviews of safety data from all parts of the study (Section 12.3.6.2). Procedural details of the IDMC structure and function, frequency of meetings, and data planned for review will be included in the IDMC Charter. The IDMC Charter will be finalized before the first subject is screened.

# 8.2 Rationale for Study Design and Study Drug Regimens

#### 8.2.1 Study Design

This Phase 2 study is the first study to assess combination therapy of VX-440 with TEZ and/or IVA in subjects with CF.

Parts 1 and 2 are designed to evaluate the safety and efficacy of the TC and to establish proof-of-concept in 2 populations of subjects defined by *CFTR* genotype: subjects heterozygous for the *F508del* mutation with a second *CFTR* allele carrying an minimal CFTR function mutation that is not expected to respond to TEZ/IVA (*F508del*/MF) (Part 1), and subjects homozygous for *F508del* (*F508del*/F508del) (Part 2) (See Section 8.2.3).

Based on in vitro data, TC is predicted to provide clinically relevant improvements in chloride transport in both populations greater than the individual compounds or any dual combinations. In Parts 1 and 2, efficacy will be evaluated through the assessment of spirometry and patient reported outcomes, and PD will be evaluated through the assessment of sweat chloride. Part 1 of the study will also obtain information regarding the exposure-response relationship (Section 12.1.2.1).

A Phase 3 study of TEZ/IVA in subjects with *F508del*/MF genotypes (Study VX14-661-107) was terminated following a planned interim futility analysis that showed that the combination of TEZ/IVA did not result in a prespecified improvement in lung function. Efficacy has not been established for a corrector, potentiator, or any corrector/potentiator combination in subjects with *F508del*/MF genotypes. Therefore, placebo is the comparator in Part 1.

A potential for benefit was demonstrated for TEZ/IVA in subjects with the *F508del/F508del* genotype in Study VX11-661-101. Therefore, TEZ/IVA is the comparator in Part 2. In addition, Part 2 will have a 4-week run-in period to establish a reliable on-treatment (TEZ/IVA) baseline for comparison to the Treatment Period, when subjects will additionally receive VX-440 or placebo.

To measure off-treatment effects, Part 1 will include a Day 43 Visit, and Part 2 will include a VX-440 (or placebo) washout period.



# 8.2.2 Study Drug Dose and Duration

#### VX-440 Dose

Part 1 will evaluate 2 dose levels of VX-440 in TC with TEZ/IVA in subjects with the F508del/MF genotype. The planned high dose of VX-440 to be evaluated as part of the TC (TC-1B-high) is 600 mg q12h which was the highest dose shown to be safe and well tolerated in TC in healthy subjects in Study 002. This dose was selected to ensure maximal clinical benefit based on the in vitro potency of VX-440 as part of the TC, while maintaining a margin of exposure relative to safety findings from nonclinical studies. The low dose (TC-1B-low) of 200 mg q12h is also predicted to provide clinical benefit based on in vitro data and was selected to provide a lower range of exposure for exposure-response analyses of safety and efficacy.

It is anticipated that differences in VX-440 PK may be observed in subjects with CF relative to healthy subjects, based on previous clinical experience with another CFTR corrector of similar dose range, LUM, where lower exposures were observed in subjects with CF relative to healthy subjects. Thus, the planned high dose of VX-440 (600 mg q12h) may result in lower exposure in

patients relative to the highest exposure evaluated in healthy subjects, if an effect similar to LUM is observed for VX-440. If VX-440 exposures in Cohort 1A are higher than that in healthy subjects at a comparable dose, then the high dose of VX-440 will be reduced from 600 mg q12h to 400 mg q12h.

Dose- and exposure-response information obtained from Part 1 (subjects with the F508del/MF genotype) is expected to be applicable to other populations with an F508del mutation, including subjects with the F508del/F508del genotype, based on similar in vitro potency for the TC in HBE cells with 1 or 2 copies of  $F508del.^8$ 

#### **TEZ Dose**

In Cohort 1A, TEZ will be administered as 100 mg qd, which is the same dose currently under evaluation in Phase 3 studies of TEZ/IVA. This dose of TEZ is appropriate for evaluation in the TC based on in vitro experiments with VX-440 which evaluated similar levels of TEZ exposure after correction for protein-binding. In Cohort 1B and Part 2, the dose of TEZ, when administered in the TC, will be 50 mg q12h so that all components of the TC are administered q12h; the total daily dose of TEZ (100 mg) will be the same as that under evaluation in Phase 3 studies of TEZ/IVA.

#### **IVA Dose**

In vitro data indicate that maintaining adequate IVA exposure in vivo will be important for maximizing efficacy of the TC. When administered in combination with VX-440 200 mg, the dose of IVA will be the same as the recommended dose for IVA monotherapy for patients aged 12 years and older (150 mg q12h). Preliminary data from Study 002 indicate that VX-440 is a moderate to strong inducer of CYP3A4. Because IVA is a sensitive CYP3A substrate, the dose of IVA will be increased from 150 mg q12h to 300 mg q12h when it is administered with VX-440 at a dose level of 600 mg q12h. These dose levels were evaluated in Study 002 and were safe and well tolerated. At these dose levels, IVA exposure was approximately 50% lower relative to IVA 150 mg q12h monotherapy based on historical data. 12 If the high dose of VX-440 is reduced to 400 mg q12h, the IVA dose will remain 300 mg q12h, as VX-440 induction is predicted to be similar in magnitude at this dose relative to 600 mg q12h. Phase 3 and postapproval data for IVA monotherapy have not revealed any systemic exposure-related safety findings and indicate a wide therapeutic margin for safety. Use of a higher IVA dose when coadministering IVA with a CYP3A inducer is consistent with the approach for combination therapy with LUM (a strong CYP3A inducer). In that combination therapy, the IVA dose is 250 mg q12h.

#### Treatment Duration

The 4-week treatment duration in Parts 1 and 2 is based on previous experience with CF correctors and potentiators in clinical studies of subjects with CF. Based on preliminary data from Studies 001 and 002, and data from previous studies of TEZ and IVA, all components of the TC reach steady-state levels of exposure by 2 to 3 weeks. In previous studies of TEZ and IVA, PD effects were observed within 4 weeks of treatment. In Study VX06-770-101, treatment with IVA for 28 days resulted in statistically significant within-group changes from baseline in ppFEV<sub>1</sub> as well as a trend toward clinically meaningful improvements in the respiratory domain of the CFQ-R; differences in biomarkers of CFTR activity (sweat chloride) between IVA and placebo groups were also demonstrated. Furthermore, in Study VX11-661-101 dose-dependent

improvements in lung function were observed for TEZ/IVA after 4 weeks of treatment, with the 2 highest dose groups showing statistically significant improvement in lung function versus placebo. In both studies, improvements in sweat chloride and ppFEV<sub>1</sub> were observed as rapidly as 3 to 7 days after the start of dosing, with most of the effect observed within 14 days. Given the increased in vitro response of the TC relative to TEZ/IVA, it is expected that the 4-week treatment duration in Parts 1 and 2 will be sufficient to observe differences between treatment arms with respect to efficacy and PD endpoints.



#### 8.2.3 Rationale for Study Population

The study will include subjects with F508del/MF and F508del/F508del genotypes based on in vitro data that indicate the potential for significant improvements in chloride transport for CF patients with 1 or 2 copies of the F508del mutation in response to treatment with TC compared to individual compounds and all dual combinations. The subjects will be evaluated by genotype in separate cohorts in Parts 1 and 2, based on the potential for differences in the magnitude of treatment response among the 2 genotype categories.

Adult subjects (age 18 years or older) will be enrolled in Parts 1 and 2. Pending demonstration of acceptable safety and the potential for benefit based on efficacy results in Part 1,

#### 8.2.4 Rationale for Study Assessments



The PD and efficacy assessments are widely accepted and generally recognized as reliable, accurate, and relevant to the study of patients in CF. All assessments,

were routinely measured in the registration studies of IVA

(Kalydeco) or LUM/IVA combination therapy (Orkambi).



#### 9 STUDY POPULATION

Eligibility will be reviewed and documented by an appropriately qualified member of the investigator's team before subjects are randomized (Parts 1 are receive TEZ/IVA in the Run-in Period (Part 2).

### 9.1 Inclusion Criteria

- 1. Subject (or subject's legally appointed and authorized representative) will sign and date an informed consent form (ICF), and, when appropriate, an assent form.
- 2. Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
- 4. Body weight  $\geq$ 35 kg.
- 5. Sweat chloride value ≥60 mmol/L from test results obtained during screening. If the value cannot be determined from the screening test, a sweat chloride value documented in the subject's medical record may be used to establish eligibility. (It is acceptable to use a sweat chloride value that was obtained before previous treatment with IVA, LUM/IVA, or an investigational CFTR modulator).
- 6. Subjects must have an eligible *CFTR* genotype as noted below. If the screening *CFTR* genotype result is not received before randomization (Parts 1 or before Day -28 (Part 2), a previous *CFTR* genotype laboratory report may be used to establish eligibility. Note: Subjects who have been randomized and whose screening genotype does not confirm study eligibility must be discontinued from the study (Section 9.5).
  - Part 1 : Heterozygous for *F508del* with a second *CFTR* allele carrying an MF mutation that is not likely to respond to TEZ and/or IVA therapy (Appendix A)
  - Part 2: Homozygous for F508del
- 7. Parts 1, 2, subjects must have an FEV₁ ≥40% and ≤90% of predicted normal for age, sex, and height (equations of the Global Lung Function Initiative [GLI])¹³ at the Screening Visit. Spirometry measurements must meet American Thoracic Society/European Respiratory Society criteria¹⁰ for acceptability and repeatability.
- 8. Stable CF disease as judged by the investigator.
- Willing to remain on a stable CF medication regimen through the planned end of treatment or, if applicable, the Safety Follow-up Visit.

#### 9.2 Exclusion Criteria

- 1. History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
- 2. History of cirrhosis with portal hypertension.
- 3. Risk factors for Torsade de Pointes, including but not limited to, history of any of the following: familial long QT syndrome, chronic hypokalemia, heart failure, left ventricular hypertrophy, chronic bradycardia, myocardial infarction, cardiomyopathy, history of arrhythmia (ventricular or atrial fibrillation), obesity, acute neurologic events (subarachnoid hemorrhage, intracranial hemorrhage, cerebrovascular accident, or intracranial trauma), or autonomic neuropathy.
- 4. History of hemolysis.
- 5. G6PD deficiency, defined as G6PD activity less than the lower limit of normal (LLN) or 70% of the mean of the LLN and the ULN, whichever is greater.
- 6. Any of the following abnormal laboratory values at screening:
  - Hemoglobin <10 g/dL
  - Total bilirubin >2 × ULN
  - Aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transpeptidase (GGT), or alkaline phosphatase (ALP) ≥3 × ULN
  - Abnormal renal function defined as glomerular filtration rate ≤50 mL/min/1.73 m<sup>2</sup>
     (calculated by the Modification of Diet in Renal Disease Study Equation)<sup>14, 15</sup> for subjects
     ≥18 years of age and ≤45 mL/min/1.73 m<sup>2</sup> (calculated by the Counahan-Barratt
     equation)<sup>16</sup> for subjects aged 12 to 17 years (inclusive)
- 7. An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before the first dose of study drug (Day 1 for Parts 1 Day -28 for Part 2).
- 8. Lung infection with organisms associated with a more rapid decline in pulmonary status (e.g., *Burkholderia cenocepacia*, *Burkholderia dolosa*, and *Mycobacterium abscessus*). For subjects who have had a history of a positive culture in the past, the investigator will apply the following criteria to establish whether the subject is free of infection with such organisms:
  - The subject has had 2 respiratory tract cultures negative for these organisms within the past 12 months, with no subsequent positive cultures.
  - These 2 respiratory tract cultures were separated by at least 3 months, and 1 of them was obtained within the past 6 months.
- 9. An acute illness not related to CF (e.g., gastroenteritis) within 14 days before the first dose of study drug (Day 1 for Parts 1 Day -28 for Part 2).

- 10. A standard digital ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec for the screening ECG, the ECG should be repeated 2 more times during the Screening Period, and the subject will be excluded if the average of the 3 QTc values is >450 msec.
- 11. History of solid organ or hematological transplantation.
- 12. History or evidence of cataract or lens opacity determined to be clinically significant by the ophthalmologist or optometrist based on the ophthalmologic examination during the Screening Period. If there is documentation of an examination meeting protocol criteria that was conducted within 3 months before the date of informed consent (or assent, when applicable), then the ophthalmologic examination does not need to be repeated during the Screening Period. This criterion does not apply to subjects with documentation of bilateral lens removal, and the ophthalmologic examination is not required for these subjects at screening.
- 13. History of alcohol or drug abuse in the past year, including but not limited to, cannabis, cocaine, and opiates, as deemed by the investigator.
- 14. Ongoing or prior participation in an investigational drug study with the exception of the following:
  - Ongoing or prior participation in an investigational study of TEZ/IVA, IVA, LUM/IVA, or other CFTR modulator. For Parts 1 a washout period of 28 days must elapse before Day 1. Subjects participating in Study 661-110 may have the Part 1 Screening Period extended by 4 weeks (Section 8.1.1.3). For Part 2, a washout period before Day -28 is not required, and subjects participating in Study 661-110 will transition directly from their prior treatment to the TEZ/IVA Run-in Period providing that they meet eligibility criteria. For all parts, subjects participating in Study 661-110 may have their screening assessments performed while continuing to participate in Study 661-110.
  - For prospective subjects with ongoing or prior participation in all other interventional studies, a washout period of 28 days or 5 terminal half-lives, whichever is longer, must elapse before screening. The duration of the elapsed time may be longer if required by local regulations.
  - Ongoing participation in a noninterventional study (including observational studies and studies requiring assessments without administration of study drug or assignment to other interventions) is permitted.
- 15. Use of commercially available CFTR modulator (e.g., Kalydeco, Orkambi) within 14 days before screening (Parts 1
- 16. Use of restricted medications as defined in Table 9-1, within the specified window before the first dose of study drug (Day 1 in Parts 1 , Day -28 in Part 2).
- 17. Pregnant or nursing females: Females of childbearing potential must have a negative pregnancy test at screening and Day 1.
- 18. The subject or a close relative of the subject is the investigator or a subinvestigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of

the study. An adult (aged 18 years or older) who is a relative of a study staff member may be randomized in the study provided that

- the adult lives independently of and does not reside with the study staff member, and
- the adult participates in the study at a site other than the site at which the family member is employed.

### 9.3 Prohibited Medications

Medications that are prohibited in this study (Screening Period through the Safety Follow-up Visit) are shown in Table 9-1. VX-440, TEZ, and IVA are metabolized extensively via CYP3A4. VX-440 is also metabolized extensively by CYP2C9 and to a lesser extent by CYP2C19. Therefore, the use of moderate and strong inducers of CYP3A or CYP2C9 and strong and moderate inhibitors of CYP3A, which have the potential to alter the exposure of VX-440, TEZ, or IVA, will be restricted in this study. Preliminary results from Study 002 indicate that VX-440 is a moderate to strong inducer of CYP3A4 at higher doses; therefore, sensitive CYP3A substrates with a narrow therapeutic index should be used with caution during the study. VX-440 was shown in vitro to be an inhibitor of the hepatic transporter organic anion transporting polypeptide 1B1 (OATP1B1). Therefore, sensitive substrates of OATP1B1, such as HMG Co-A Reductase Inhibitors (i.e., "statins"), are restricted during treatment with VX-440 or placebo. As VX-440 has demonstrated the potential for inhibition of CYP2C9 in vitro, warfarin is also prohibited during treatment with VX-440 or placebo.

A non-exhaustive list of study prohibitions and cautions for medication will be provided in the Study Reference Manual.

Table 9-1 Prohibited Medications

| | Timing of Re | estriction |
|---|---|---|
| Medication | Start of Restriction | End of Restriction |
| Moderate and strong CYP3A or CYP2C9 inducers | None allowed within 14 days before the first dose of the study drug on Day 1 (Parts 1 Day -28 (Part 2) | None allowed through the Safety<br>Follow-up Visit |
| Moderate and strong CYP3A inhibitors (except ciprofloxacin) | None allowed within 14 days before the first dose of the study drug on Day 1 (Parts 1 Day -28 (Part 2) | None allowed through the Safety<br>Follow-up Visit |
| Sensitive OATP1B1 substrates | None allowed within 14 days before the first dose of VX-440 or placebo on Day 1 | None allowed until after last dose of VX-440 or placebo |
| Warfarin | None allowed within 14 days before the first dose of VX-440 or placebo on Day 1 | None allowed until after last dose of VX-440 or placebo |
| Commercially available CFTR modulators (e.g., | Parts 1 None allowed within 14 days before screening | Parts 1 None allowed through the Safety Follow-up Visit |
| Kalydeco, Orkambi) | Part 2: None allowed from the start of the Run-in Period | Part 2: None allowed through end of the Washout Period |

CFTR: Cystic fibrosis transmembrane conductance regulator; CYP: cytochrome P450; OATP1B1: organic anion transporting polypeptide 1B1

Note: The use of restricted medication by subjects with medical needs will be addressed on a case-by-case basis with the medical monitor.

#### 9.4 Prior and Concomitant Medications

Information regarding all prior and concomitant medications, including the subject's CF medications, other medications, and herbal and naturopathic remedies administered from 28 days before the Screening Visit through the Safety Follow-up Visit, if applicable, will be recorded in each subject's source documents. For subjects who are screened but are not subsequently randomized in the study, details of prior medication will only be documented in the subjects' source documents.

- Subjects must remain on a stable medication (and supplement) regimen for their CF from 28 days before Day 1 through the Safety Follow-up Visit. Stable medication regimen is defined as the current medication regimen for CF that subjects have been following for at least 28 days before Day 1. Subjects must not initiate long-term treatment with new medication from 28 days before Day 1 through the Safety Follow-up Visit unless discussed and approved by the medical monitor. Guidelines for stable medication regimens for CF are as follows:
  - Subjects who are taking daily inhaled tobramycin or other chronically inhaled antibiotics should remain on that regimen throughout the study.
  - Subjects who cycle onto and off of an inhaled antibiotic should continue on their prior schedule. The timing of the first dose of study drug on Day 1 should be synchronized as closely as possible (and not more than ± 3 days) to the first day in the cycle onto the inhaled antibiotic.
  - Subjects who alternate between 2 different inhaled antibiotics should remain on the same cycling schedule during the study. The timing of the first dose of study drug on Day 1 should be synchronized as closely as possible (and not more than ± 3 days) to the first day in the cycle onto 1 of the inhaled antibiotics.
- Subjects may receive doses of prednisone of up to 10 mg/day or equivalent (chronically) or prednisone 60 mg qd for up to 5 days without prior approval of the medical monitor.
- Information about bronchodilator use during the study will be collected and documented.
   Subjects who are using a bronchodilator must have their spirometry assessments performed according to the guidelines provided in Section 11.6.1.

### 9.5 Removal of Subjects

Subjects may withdraw from the study at any time at their own request. Subjects may be withdrawn from study drug treatment at any time at the discretion of the investigator or Vertex for safety, behavior, noncompliance with study procedures, or administrative reasons. If a subject has been withdrawn from study drug treatment, the subject will continue to be followed, provided the subject has not withdrawn consent.

Subjects who have been randomized and whose screening *CFTR* genotype does not confirm study eligibility must be discontinued from the study, even if a previous *CFTR* genotype laboratory report was used to establish eligibility.

If a subject does not return for a scheduled visit, reasonable effort will be made to contact the subject. In any circumstance, reasonable effort will be made to document subject outcome. The investigator will inquire about the reason for withdrawal, request that the subject return all unused investigational product(s), request that the subject return for a Safety Follow-up Visit, if applicable (see Section 8.1.6), and follow up with the subject regarding any unresolved AEs.

If the subject withdraws consent for the study, no further evaluations will be performed and no additional data will be collected. Vertex may retain and continue to use any data collected before such withdrawal of consent.

### 9.6 Replacement of Subjects

Subjects who withdraw or are withdrawn before the first dose of study drug on Day 1 may be replaced.

Subjects who withdraw or are withdrawn for nonsafety reasons during the study drug treatment period may be replaced at Vertex's discretion.

### 10 STUDY DRUG ADMINISTRATION AND MANAGEMENT

Study drug refers to VX-440, TEZ/IVA, TEZ, IVA, and their matching placebos.

## 10.1 Preparation and Dispensing

Study drug may be dispensed only under the supervision of the investigator or an authorized designee and only for administration to the study subjects.

#### 10.2 Administration

Study drug will be administered orally. Subjects will receive the same number of tablets each day to maintain the blind. Additional information is provided in the Pharmacy Manual.

Study drug will be administered with a fat-containing meal or snack, such as a standard "CF" high-fat, high-calorie meal or snack or a standard meal, according to the following guidelines:

- 1. It is recommended that the dose be taken within 30 minutes of the start of the meal or snack.
- 2. Study drug will be administered q12h ( $\pm$  2 hours). For each subject, all doses of study drugs will be taken at approximately the same time each day. For example, the morning dose could be taken at 08:00 every morning and the evening dose could be taken at 20:00 every evening throughout the study.
- 3. The date, amount taken, and time of study drug administration, including whether food was taken with each dose, will be recorded for the 2 doses before PK sample collection and the dose received on the morning of PK sample collection.
- 4. On days of scheduled visits, the morning dose of study drug will be administered at the site after predose assessments have been completed. The meal or snack will be provided by the site for the morning dose of study drug.

- 5. If a subject's scheduled visit is to occur in the afternoon, the following guidelines must be used:
  - If the dose in the clinic will be within 6 hours of the subject's scheduled morning dose, the subject should withhold their morning dose of study drug and the morning dose will be administered in the clinic.
  - If the dose in the clinic will be more than 6 hours after the subject's scheduled morning dose, the subject should take the morning dose at home and the evening dose will be administered in the clinic. In this event, all assessments will be collected relative to the evening dose.
- 6. Subjects will be instructed to bring all used and unused study drug to the site; study drug will be dispensed at each visit, as appropriate.

#### 10.2.1 Missed Doses

If a subject misses a dose and recalls the missed dose within 6 hours, the subject should take his/her dose with food. If more than 6 hours have elapsed after his/her usual dosing time, the subject should skip that dose and resume his/her normal schedule for the following dose. For example,

- if the morning dose of study drug should have been taken at approximately 08:00, and the subject remembers at 12:00 that he/she forgot to take his/her dose, he/she should take the dose with food as soon as possible.
- if the morning dose of study drug should have been taken at approximately 08:00, and more than 6 hours have elapsed beyond the scheduled dosing time (i.e., the time is past 14:00), the subject would resume dosing with the evening dose at approximately 20:00.

# 10.3 Method of Assigning Subjects to Treatment Groups

Treatment arms, randomization ratios, and stratification factors for each part are described in Table 8-1. An interactive web response system (IWRS) will be used to assign subjects to treatment. The randomization code list will be produced by Vertex Biometrics or a qualified randomization vendor.

# 10.4 Study Drug Interruption and Stopping Rules

Subjects with new treatment-emergent ALT or AST elevations of  $>3 \times ULN$ , or total bilirubin  $>2 \times ULN$ , must be followed closely, including confirmatory testing performed by the central laboratory within 48 to 72 hours of the initial finding and subsequent close monitoring of ALT, AST, and bilirubin levels, as clinically indicated.

If a subject cannot return to the site for confirmatory testing, a local laboratory may be used. Local laboratory results must be reported immediately to the medical monitor, and the subject must have the tests repeated and sent to the central laboratory as soon as possible (ideally within 48 to 72 hours).

Study drug administration <u>must be interrupted</u> immediately (prior to confirmatory testing), and the medical monitor must be notified, if any of the following criteria are met:

- ALT or AST >8 × ULN
- ALT or AST >5 × ULN for more than 2 weeks

- ALT or AST >3 × ULN, in association with total bilirubin >2 × ULN and/or clinical jaundice
- Indirect bilirubin >2 × ULN (defined as ULN for total bilirubin minus ULN for direct bilirubin)

A thorough investigation of potential causes should be conducted, and the subject should be followed closely for clinical progression.

Study drug administration **must be discontinued**, if either of the following criteria is met:

- Subsequent ALT or AST values confirm the initial elevation that satisfied the interruption
  rule (above), and no convincing alternative etiology (e.g., acetaminophen use, viral hepatitis,
  or alcohol ingestion) is identified, regardless of whether transaminase levels have improved
- Indirect bilirubin >2 × ULN (defined as ULN for total bilirubin minus ULN for direct bilirubin), in association with decreased haptoglobin

If an alternative, reversible cause of transaminase elevation and/or increased bilirubin or clinical jaundice has been identified, study drug administration may be resumed once transaminases or bilirubin return to baseline or are  $\leq 2 \times ULN$ , whichever is higher. Approval of the medical monitor is required before resumption of study drug. Upon resumption of study drug, transaminases and bilirubin should be assessed weekly for 4 weeks. If a protocol-defined transaminase or bilirubin elevation interruption threshold recurs within 4 weeks of rechallenge with the study drug (with confirmation of the initial elevation by repeat testing within 48 to 72 hours), then the study drug must be permanently discontinued, regardless of the presumed etiology.

All subjects in whom treatment is discontinued for elevated transaminases and/or bilirubin should have these levels monitored closely until levels normalize or return to baseline.

### 10.5 Packaging and Labeling

Study drug tablets will be supplied in blister cards by Vertex. Study drug labeling will be in compliance with applicable local and national regulations. Additional details regarding packaging, labeling, and dispensing for study drug will be included in the Pharmacy Manual.

### 10.6 Study Drug Supply, Storage, and Handling

VX-440 (200 mg) and matching placebo will be supplied as tablets of similar size and appearance containing 200 mg VX-440 and 0 mg VX-440, respectively.

TEZ/IVA (100 mg/150 mg) and matching placebo will be supplied as light yellow film-coated tablets of similar size and appearance containing 100 mg TEZ/150 mg IVA and 0 mg TEZ/0 mg IVA, respectively.

TEZ (50 mg) and matching placebo will be supplied as white tablets of similar size and appearance containing 50 mg TEZ and 0 mg TEZ, respectively.

IVA (150 mg) and matching placebo will be supplied as light blue film-coated tablets of similar size and appearance containing 150 mg IVA and 0 mg IVA, respectively.

Blister cards must be stored under conditions noted in Table 10-1 and in the Pharmacy Manual. The investigator, or an authorized designee (e.g., a licensed pharmacist), will ensure that all investigational product is stored in a secured area, under recommended storage conditions, and in

accordance with applicable regulatory requirements. To ensure adequate records, all study drugs will be accounted for via the drug accountability forms as instructed by Vertex.

Table 10-1 Study Drug

| | Strength/Formulation/ | | |
|---|---|---|---|
| Drug Name | Route | Dosage | Storage Condition |
| VX-440 | 200-mg tablet, oral | 200 mg q12h<br>600 mg q12h<br>(planned) | ≤25°C (77°F) with<br>excursions to 30°C (86°F) |
| VX-440-matching placebo | 0-mg tablet, oral | 0 mg q12h | ≤25°C (77°F) with excursions to 30°C (86°F) |
| TEZ/IVA fixed-dose | 100-mg/150-mg tablet; oral | 100 mg/150 mg qd<br>(morning dose) | ≤25°C (77°F) with excursions to 30°C (86°F) |
| TEZ/IVA-matching placebo | 0-mg/0-mg tablet; oral | 0 mg/0 mg qd<br>(morning dose) | ≤25°C (77°F) with excursions to 30°C (86°F) |
| TEZ | 50-mg tablet, oral | 50 mg q12h | ≤25°C (77°F) with excursions to 30°C (86°F). |
| TEZ-matching placebo | 0-mg tablet, oral | 0 mg q12h | ≤25°C (77°F) with excursions to 30°C (86°F) |
| IVA | 150-mg tablet, oral | 150 mg qd<br>(evening dose)<br>150 mg q12h | ≤25°C (77°F) with<br>excursions to 30°C (86°F) |
| IVA-matching placebo | 0-mg tablet, oral | 0 mg qd<br>(evening dose)<br>0 mg q12h | ≤25°C (77°F) with excursions to 30°C (86°F) |

IVA: ivacaftor; q12h: every 12 hours; qd: daily; TBD: to be determined

# 10.7 Drug Accountability

The pharmacist or designated study site staff will maintain information regarding the dates and amounts of study drug received; study drug dispensed to the subjects; and study drug returned by the subjects. Subjects will be instructed to return all used and unused materials associated with the study drug to the site. These materials will be retained at the site according to instructions provided by Vertex or its designee until inventoried by the study monitor. The study monitor will review study drug records and inventory throughout the study.

# 10.8 Disposal, Return, or Retention of Unused Drug

The study site staff or pharmacy personnel will retain all materials returned by the subjects until the study monitor has performed drug accountability. At the end of the study, the study monitor will provide instructions as to the disposition of any unused investigational product. If the study monitor authorizes destruction at the study site, the investigator will ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Vertex. Destruction will be adequately documented.

# 10.9 Compliance

To ensure treatment compliance, the investigator or designee will supervise all study drug dosing that occurs at the site. At each visit, site personnel will review that the subject is compliant with study drug dosing and remind the subject of study drug dosing requirements. Compliance will also be assessed by ongoing study drug count.

If a subject demonstrates continued noncompliance of study drug dosing despite educational efforts, the investigator will contact the medical monitor to discuss discontinuing the subject from the study.

### 10.10 Blinding and Unblinding

This will be a double-blind study.

# 10.10.1 Blinding

All subjects, site personnel (including the investigator, the site monitor, and the study team), and the Vertex study team will be blinded to the treatment codes with the exception of the following:

- Any site personnel for whom this information is important to ensure the safety of the subject in the event of a life-threatening medical emergency
- Any site personnel for whom this information is important to ensure the safety of the subject and her fetus in the event of a pregnancy
- Vertex Global Patient Safety (GPS) and Regulatory Affairs personnel to satisfy serious adverse event (SAE) processing and reporting regulations
- Unblinded statistician preparing the final (production) randomization list who is not part of the study team
- Vertex IWRS Manager
- Vertex Clinical Supply Chain
- IDMC
- Vendor preparing the unblinded analysis for the ongoing reviews of efficacy and safety data, and the IDMC
- Vendor analyzing PK samples
- Vertex Modeling and Simulation personnel or vendor conducting the population PK and PK/PD analyses
- Vertex medical monitor may, for matters relating to safety concerns, unblind individual subjects at any time

Vertex Drug Metabolism and Pharmacokinetics laboratory personnel will not be involved in the conduct of the study and will be unblinded to the bioanalysis results but will remain blinded to subject number and treatment assignment.

<u>Spirometry and Sweat Chloride Data Blinding</u>: During the conduct of the study, the Vertex study team will not have access to the spirometry or sweat chloride results after the morning dose on Day 1. Furthermore, sites, subjects, and their parents/caregivers/companions should not be

informed of their study-related spirometry and sweat chloride results during the Treatment Period regardless of whether the subject has prematurely discontinued treatment.

A limited Vertex team will be unblinded and have access to safety, efficacy, and PD data for the purpose of conducting ongoing reviews of safety and efficacy data for planning and enabling clinical development, regulatory, and chemistry, manufacturing, and controls (CMC) decisions. Members of the limited unblinded Vertex team will not be part of the Vertex study team and will not be involved in or influence the conduct of the study.

The Vertex study team and lead investigator(s) will conduct a blinded review of all available safety and PK data after all Cohort 1A subjects complete the Day 15 Visit. The Vertex study team will not have access to unblinded data from ongoing reviews by the limited Vertex team.

After all subjects within Parts 1 and 2 have completed the Safety Follow-up Visit, results from each part will be unblinded for full review by the Vertex study team (Section 12.3.6.1).

# 10.10.2 Unblinding

At the initiation of the study, the study site will be instructed on the method for breaking the blind. The unblinding method will be either a manual or electronic process.

Unblinding of the individual subject's treatment by the investigator will be limited to medical emergencies or urgent clinical situations in which knowledge of the subject's study treatment is necessary for clinical management. In such cases, investigators will use their best judgment as to whether to unblind without first attempting to contact the medical monitor to discuss and agree to the need for unblinding. If investigators deem it not necessary to unblind immediately, they will first attempt to contact the medical monitor to discuss and agree to the need for unblinding. If investigators have tried but are unable to reach the medical monitor, they will use their best judgment, based on the nature and urgency of the clinical situation, and may proceed with unblinding without having successfully reached and discussed the situation with the medical monitor.

Contact information for the medical monitor (or appropriate backup) will be provided in a separate document.

In addition, the Vertex Medical Information Call Center ( ) will answer calls 24 hours a day, 7 days a week, 365 days of the year, and will triage these calls to the study medical monitor or appropriate backup.

If a subject's treatment assignment has been unblinded for a medical emergency or urgent clinical situation, the medical monitor will be notified within 24 hours of the unblinding event. The reason and the date of the unblinding will be documented clearly in the subject's study file. Information about the treatment assignment obtained from the unblinding will be maintained in a secure location with controlled access and will not be shared with the sponsor (Vertex), contract research organization (CRO), or any site personnel (other than the physician treating the subject). In addition, the investigator will consider whether the clinical event that prompted unblinding will be considered an SAE, according to the regulatory definitions or criteria for SAEs, and if so, submit an SAE report to Vertex GPS or designee, per Section 13.1.2.

Vertex GPS or designee will also unblind any SAE reports in compliance with regulatory reporting requirements. In addition, Vertex may, for matters relating to safety concerns, unblind individual subjects at any time.

#### 11 ASSESSMENTS

### 11.1 Timing of Assessments

The CFQ-R assessment must be completed before any other assessment at the clinic visits when it is required. For remaining assessments, assessments may be performed in any order when more than 1 assessment is required at a particular time point.



### 11.2 Subject and Disease Characteristics

Subject and disease characteristics include the following: demographics, medical history, height, and weight.

Medical history will be elicited from each subject and extracted from medical records during screening. Based on the medical history, the subject will be assessed for any disqualifying medical conditions as specified in the inclusion and exclusion criteria. The medical history shall include a complete review of systems, past medical and surgical histories, and any allergies.

#### 11.3 Pharmacokinetics

# 11.3.1 Blood Sampling

Blood samples will be collected as shown in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2), for the determination of plasma concentrations of VX-440, TEZ, M1-TEZ, IVA, and M1-IVA.

All efforts will be made to obtain the PK samples at the exact nominal time relative to dosing. Acceptable windows for sampling times are shown in Table 11-1. Samples collected outside of these acceptable windows will be considered protocol deviations.

Table 11-1 Acceptable Pharmacokinetic Sampling Windows

| Sampling Time | Time From Scheduled Sampling Allowed |
|---|---|
| Predose | -60 minutes |
| From 0.25 up to ≤8 hours after study drug dosing | ± 15 minutes |

For each visit with a PK blood draw, a record of study drug administration will be collected as described in Section 10.2. The collection date and exact time that each PK blood sample is drawn will also be recorded.

Samples from the PK sampling will be kept frozen by Vertex or its designee until all analyses have been completed and then disposed of according to Vertex or designee standard operating procedures.

Plasma concentration samples collected from subjects treated with placebo will not be routinely analyzed.

# 11.3.2 Processing and Handling of Pharmacokinetic Samples

Detailed procedures for the collection of blood samples and further procedures for processing and handling of samples for PK analysis will be provided in the PK Sample Handling Guidelines. The shipment address and assay laboratory contact information will be provided to the investigational site before initiation of the study.

# 11.3.3 Bioanalysis

Samples will be analyzed using 1 or more validated analytical methods in compliance with Vertex or designee standard operating procedures. A description of the assay and validation data will be provided in separate reports.

# 11.4 Pharmacodynamics

### 11.4.1 Sweat Chloride

The sweat chloride test is a standard diagnostic tool for CF, serving as a biomarker of CFTR activity. Collection of sweat samples will be performed at visits specified in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2), using an approved collection device. At each time point, 2 samples will be collected, 1 from each arm (left and right). Sweat samples will be sent to a central laboratory for testing and interpretation of results. Individual sweat chloride test results will not be disclosed to the study sites with the exception of the screening values. Specific instructions for collection, handling, processing, and shipping of sweat chloride samples to the central laboratory will be provided separately.

Subjects and their parents/caregivers/companions should not be informed of their study-related sweat chloride results during the Treatment Period, regardless of whether the subject prematurely discontinues treatment.



### 11.6 Efficacy

### 11.6.1 Spirometry

Spirometry will be performed according to the American Thoracic Society Guidelines/European Respiratory Society Guidelines<sup>10</sup> at the time points noted in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2), and according to the additional guidelines that follow.

Pre-bronchodilator spirometry is defined as spirometry testing performed for subjects who have

- withheld their short-acting bronchodilators (e.g., albuterol) or anticholinergic (e.g., ipratropium bromide [Atrovent<sup>®</sup>]) for more than 4 hours before the spirometry assessment;
- withheld their long-acting bronchodilator (e.g., salmeterol) for more than 12 hours before the spirometry assessment; and
- withheld their once-daily, long-acting bronchodilator (e.g., tiotropium bromide [Spiriva®]) for more than 24 hours before the spirometry assessment.

During the Screening Period, spirometry assessments may be performed pre- or post-bronchodilators. At all other visits, all spirometry assessments should be performed "pre-bronchodilator". During the Treatment Period, spirometry assessments must be performed before the morning dose of study drugs at approximately the same time at each visit. Postdose spirometry assessments will be performed as noted in Table 3-1, Table 3-2, Table 3-3,

In the event that a subject forgets to withhold bronchodilator(s), spirometry should be performed according to the following:

- If a subject's Day 1 spirometry assessment is pre-bronchodilator, but, on a subsequent visit, the subject forgets to withhold bronchodilator use, a post-bronchodilator spirometry assessment will be obtained for that visit only, and the visit will not be rescheduled.
- If, on Day 1, the subject forgets to withhold his/her dose of bronchodilator, spirometry should be performed post-bronchodilator, and all subsequent spirometric measurements (according to the schedule of assessments detailed in Table 3-1, Table 3-2, Table 3-3, should be performed post-bronchodilator.
- Each spirometry assessment will be recorded in the source documents as pre- or post-bronchodilator.

If more than 1 spirometry assessment is required at a visit, bronchodilators will be withheld until completion of the last scheduled spirometry assessment.

All sites will be provided with spirometers to be used for all study assessments. Spirometry data will be transmitted to a centralized spirometry service for quality review.

Subjects and their parents/caregivers/companions should not be informed of their study-related spirometry results during the Treatment Period, regardless of whether the subject prematurely discontinues treatment.

The measured spirometric values listed below will be converted to percent predicted values using the standards of GLI.<sup>13</sup>



# 11.6.2 Height and Weight

Height and weight will be measured with shoes off at time points noted in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2),

# 11.6.3 Cystic Fibrosis Questionnaire-Revised

Subjects will be asked to complete the CFQ-R in their native language, if validated translations are available. <sup>17, 18</sup> The CFQ-R will be completed before any other study assessments are performed at the visits noted in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2),

The questionnaires

provide information about demographics; general quality of life, school, work, or daily activities; and symptom difficulties (pertaining to CF). Copies of the CFQ-R used in this study will be provided in the Study Reference Manual. Validated translations of the CFQ-R, if available, will be provided for participating centers in non-English-speaking countries.<sup>19, 20</sup>



# 11.7 Safety

Safety evaluations will include AEs, clinical laboratory assessments, ECGs, clinical evaluation of vital signs, pulse oximetry, PEs, and ophthalmologic examinations.

#### 11.7.1 Adverse Events

All AEs will be assessed, documented, and reported in accordance with ICH GCP guidelines. Section 13.1 outlines the definitions, collection periods, criteria, and procedures for documenting, grading, and reporting AEs. A separate document that details AE case report form (CRF) completion guidelines for investigators as well as training will be provided.

# 11.7.2 Clinical Laboratory Assessments

Blood and urine samples will be analyzed at a central laboratory, with the exception of the urine pregnancy tests which will be performed and analyzed at the site. Fasting is not required. On Day 1, blood samples will be collected before the first dose of the study drug.

Blood and urine samples for clinical laboratory assessments will be collected as shown in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2), Laboratory test results that are abnormal and considered clinically significant will be reported as AEs.

The safety laboratory test panels are shown in Table 11-2.

| Serum Chemistry | <b>Hematology</b> <sup>a</sup> | Urinalysis <sup>b</sup> |
|---|---|---|
| Serum Chemistry Glucose Blood urea nitrogen Creatinine Sodium Potassium Calcium Chloride Magnesium Bicarbonate | Hemoglobin Erythrocytes Mean corpuscular hemoglobin Mean corpuscular hemoglobin concentration Mean corpuscular volume Reticulocytes Platelets Leukocytes | Urinalysis <sup>b</sup> Leukocyte esterase Nitrite Urobilinogen Urine protein pH Urine blood Specific gravity Urine ketones Urine bilirubin |
| Inorganic phosphate Total bilirubin Direct bilirubin Alkaline phosphatase Aspartate aminotransferase Alanine aminotransferase | Differential (absolute and percent): Eosinophils Basophils Neutrophils Lymphocytes Monocytes | Urine glucose |
| Lactate dehydrogenase Gamma-glutamyl transpeptidase Total protein Albumin Amylase Lipase Haptoglobin <sup>c</sup> | Activated partial thromboplastin time Prothrombin time Prothrombin time International Normalized Ratio | |

Table 11-2 Safety Laboratory Test Panels

Pregnancy (β-human chorionic gonadotropin) Tests for Females of Childbearing Potential: Serum samples will be obtained as specified in Table 3-1, Table 3-2, Table 3-3, and analyzed at the central laboratory. Urine pregnancy tests will be performed at the site as specified in Table 3-1, Table 3-2, Table 3-3, The urine pregnancy test on Day 1 must be negative before the first dose of study drug. Additional urine pregnancy tests may be required according to local regulations and/or requirements.

<u>Follicle-stimulating Hormone (Screening Period only)</u>: Blood sample for FSH will be measured for any suspected postmenopausal female with at least 12 months of continuous spontaneous amenorrhea. Serum FSH levels must be within the postmenopausal reference range of the performing laboratory to be considered postmenopausal.

<u>CFTR</u> genotype (Screening Period only): CFTR genotyping will be performed for all subjects. If the screening CFTR genotype result is not received before randomization, a previous CFTR genotype laboratory report may be used to establish eligibility. Subjects who have been randomized and whose screening genotype does not confirm study eligibility must be discontinued from the study (Section 9.5).

<u>G6PD Activity Test (Screening Period only)</u>: A single blood sample will be collected for the G6PD activity test, which will be performed in an established laboratory that runs the assay routinely.

Blood smears will be saved for future evaluation, if needed.

If urine is positive for leukocyte esterase, nitrite, protein, or blood, microscopic examination of urine will be performed for leukocytes, erythrocytes, crystals, bacteria, and casts.

<sup>&</sup>lt;sup>c</sup> Haptoglobin will be analyzed only if there is evidence of possible hemolysis.

<u>Additional Evaluations:</u> Additional clinical laboratory evaluations will be performed at other times if judged to be clinically appropriate.

For purposes of study conduct, only laboratory tests done in the central laboratory may be used. Local laboratories may be used at the discretion of the local investigator for management of urgent medical issues. If a local laboratory test value is found to be abnormal and clinically significant, it will be verified by the central laboratory as soon as possible after the investigator becomes aware of the abnormal result. If it is not possible to send a timely specimen to the central laboratory (e.g., the subject was hospitalized elsewhere), the investigator may base the assessment of an AE on the local laboratory value.

# 11.7.3 Physical Examinations and Vital Signs

A PE of all body systems and vital signs assessment will be performed at screening and select study visits (see Table 3-1, Table 3-2, Table 3-3, At other visits, symptom-directed PEs and symptom-directed vital sign assessments can be performed at the discretion of the investigator or healthcare provider.

A complete PE includes a review of the following systems: head/neck/thyroid; eyes/ears/nose/throat (EENT); respiratory; cardiovascular; lymph nodes; abdomen; skin; musculoskeletal; and neurological. Breast, anorectal, and genital examinations will be performed when medically indicated. After screening, any clinically significant abnormal findings in PEs will be reported as AEs.

The abbreviated PE will include an assessment of the following body systems: EENT, cardiovascular system, respiratory system, abdomen, and skin.

Vital signs include blood pressure (systolic and diastolic), temperature (oral), pulse rate, and respiration rate. These will be assessed following at least a 5-minute rest in the seated position.

# 11.7.4 Pulse Oximetry

Arterial oxygen saturation by pulse oximetry will be measured at visits specified in Table 3-1 (Part 1 Cohort 1A), Table 3-2 (Part 1 Cohort 1B), Table 3-3 (Part 2), This will be assessed following at least a 5-minute rest (seated) and before study drug dosing. At visits when study drug is taken at the site, pulse oximetry will be collected before the morning dose. This is a noninvasive measure of oxygen delivery to the tissues and has been correlated with clinical status and lung function.

### 11.7.5 Electrocardiograms

Standard 12-lead ECGs will be performed using a machine with printout according to the Schedule of Assessments (Table 3-1 [Part 1 Cohort 1A], Table 3-2 [Part 1 Cohort 1B], Table 3-3 [Part 2], Additional standard 12-lead ECGs will be performed at any other time if clinically indicated.

The subject will be instructed to rest in the seated position for at least 5 minutes before having an ECG performed.

The ECG traces will be manually read at the study site at the Screening Visit and Safety Follow-up Visit. A printout of the ECG traces will be made for safety review by the investigator and maintained with source documentation. Clinically significant ECG abnormalities occurring during the study through the Safety Follow-up Visit will be recorded as AEs.

To ensure safety of the subjects, a qualified individual at the study site will make comparisons to baseline measurements. If the QTcF is increased by >45 msec from the baseline or an absolute QTcF value is ≥500 msec for any scheduled ECG, 2 additional ECGs will be performed approximately 2 to 4 minutes apart to confirm the original measurement. If either of the QTcF values from these repeated ECGs remains above the threshold value (>45 msec from baseline or ≥500 msec), a single ECG will be repeated at least hourly until QTcF values from 2 successive ECGs fall below the threshold value that triggered the repeat measurement. Further details pertaining to ECGs will be provided to sites in a separate document (ECG Manual).

### 11.7.6 Ophthalmologic Examination

Subjects will undergo an ophthalmologic examination performed by a licensed ophthalmologist or optometrist as noted in Table 3-1, Table 3-2, Table 3-3, which includes

- measurement of best corrected distance visual acuity of each eye; and
- pharmacologically dilated examination of the lens with a slit lamp.

The screening ophthalmologic examination must be completed and the results reviewed before randomization. This examination does not have to be performed if there is documentation of an examination that met protocol criteria and was within 3 months before the date of informed consent (or assent, when applicable) or if there is documentation of bilateral lens removal for the subject.

If a cataract or lens opacity is identified and determined to be clinically significant by the ophthalmologist or optometrist at the screening examination, the subject must not be randomized. If a cataract or lens opacity is identified and determined to be clinically significant by the ophthalmologist or optometrist after dosing, the subject will be notified. After discussion with the principal investigator and in collaboration with the medical monitor, the subject may elect to continue or discontinue study drug treatment. If the subject discontinues study drug treatment, the subject should complete the ETT and Safety Follow-up Visit. If the subject continues study drug treatment, more frequent ophthalmologic monitoring should be considered.

Additional ophthalmologic examinations may be conducted at the discretion of the investigator. The medical monitor should be notified of any additional ophthalmologic examinations and their results.

In addition, at screening, the following history will be obtained and documented for all subjects:

- history of steroid use
- history of trauma to the eye
- any family history of glaucoma, congenital cataracts, or cataracts arising later in life

# 11.7.7 Contraception and Pregnancy

The effects of VX-440 monotherapy or in dual or triple combination with TEZ and IVA on conception, pregnancy, and lactation in humans are not known. VX-440, TEZ, and IVA did not show genotoxic potential in a standard battery of in vitro (Ames test, Chinese hamster ovary cell chromosomal aberration) and in vivo (mouse micronucleus) studies. TEZ and IVA were each found to be nonteratogenic in embryo-fetal developmental toxicity studies in rats and rabbits. 11,12

In the embryo-fetal developmental toxicity studies, VX-440 was found to be nonteratogenic in rats; however, it demonstrated teratogenicity in rabbits.<sup>9,23</sup>

Based on these findings and following the recommendations outlined by the Heads of Medicines Agencies Clinical Trial Facilitation Group,<sup>24</sup> male subjects with female partners of childbearing potential must use a condom to avoid exposure of a potential embryo or fetus to study drug via the seminal fluid. Female subjects who are of childbearing potential will be required to use highly effective methods of contraception with low user dependency. Based on the potential for CYP induction by VX-440, hormonal methods of contraception will not be considered acceptable methods for female subjects of childbearing potential. Pregnancy testing will be performed at monthly intervals.

## 11.7.7.1 Contraception

Study participation requires compliance with the contraceptive requirements outlined in Table 11-3

**Table 11-3** Contraceptive Requirements

| Table 11-3 | Contraceptive Requirements |
|---|---|
| Male subjects <sup>a</sup> | <ul> <li>A male subject with a female partner of childbearing potential<sup>b</sup> must use a condom<br/>to avoid exposure of a potential embryo or fetus to study drug via the seminal<br/>fluid. This is required during the period starting from the first dose of study drug<br/>until 7 days after the last dose of study drug.</li> </ul> |
| Female subjects | At least 1 of the following methods must be used: |
| | <ul> <li>Continuous use of a non-hormone-releasing intrauterine device for at least 90 days<br/>before the first dose of study drug, and until 7 days after the last dose of study drug</li> </ul> |
| | <ul> <li>Bilateral tubal occlusion (e.g., ligation) in place at least 6 months before the first<br/>dose of study drug</li> </ul> |
| | <ul> <li>Postmenopausal state (defined as amenorrheic for at least 12 consecutive months<br/>and a serum FSH level within the laboratory's reference range for postmenopausal<br/>females)</li> </ul> |
| | <ul> <li>Documented hysterectomy or bilateral oophorectomy/salpingo-oophorectomy</li> </ul> |
| | <ul> <li>Male partner is infertile (e.g., bilateral orchiectomy)</li> </ul> |
| | <ul> <li>Male partner has vasectomy at least 6 months before the first dose of study drug,<br/>with a documented negative postvasectomy semen analysis for sperm</li> </ul> |

- In addition to the male condom, other methods of contraception may be used by male subjects and their female partners of childbearing potential, with the exception of female condom due to risk of tearing.
- Female partners of nonchildbearing potential must either be postmenopausal (defined as amenorrheic for at least 12 consecutive months) or have had a hysterectomy or bilateral oophorectomy/salpino-oophorectomy.
- Considered an acceptable method for female study subjects because of the potential for a drug-drug interaction with VX-440 resulting in reduced exposure and contraception failure; however, female subjects are not required to discontinue their use of hormonal contraceptives as long as they agree to use at least 1 of the methods listed above.

#### Additional notes:

• During the course of the study, if a change in a female subject's sexual partner leads to inability to comply with the requirements outlined in Table 11-3, the subject must immediately discontinue study drug and not engage in sexual intercourse with the new partner until 7 days after the last dose of study drug.

- Male subjects must not donate sperm during the period starting from the first dose of study drug until 7 days after the last dose of study drug.
- Female subjects should not nurse a child during the period starting from the first dose of study drug until 7 days after the last dose of study drug.

### 11.7.7.2 **Pregnancy**

Subjects will be counseled to inform the investigator of any pregnancy that occurs during study treatment and for 90 days after the last dose of study drug.

If a female subject or the female partner of a male subject becomes pregnant while participating in the study, study drug will be permanently discontinued immediately. The investigator will notify the medical monitor and Vertex GPS within 24 hours of the site's knowledge of the subject's (or partner's) pregnancy using the Pregnancy Information Collection Form.

If confirmed to be on active drug, the subject or partner will be followed until the end of the pregnancy and the infant will be followed for 1 year after the birth, provided informed consent is obtained. A separate ICF will be provided to explain these follow-up activities. Pregnancy itself does not constitute an AE.

### 12 STATISTICAL AND ANALYTICAL PLANS

### 12.1 Sample Size and Power

### 12.1.1 Primary Objectives

The primary objectives of the study are the evaluation of safety and tolerability, and efficacy of VX-440 in TC with TEZ/IVA (all parts). The sample size calculations described below are deemed adequate to evaluate the objectives of the study, based on clinical and statistical considerations.

# 12.1.1.1 Safety and Tolerability

The primary safety endpoint is the incidence of AEs. Approximately 198 subjects will be enrolled in the study with approximately 160 subjects receiving VX-440 or triple combination with IVA and/or TEZ. The sample size for each treatment group will provide sufficient data for a descriptive analysis of AEs. Table 12-1 provides the probability of observing an AE in at least 1 subject based on sample sizes ranging from 10 to 50 subjects per treatment group and AE incidences ranging from 5% to 15%. The probability calculations are based on a binomial model using the probability calculator in the PASS software package (Version 11.0).

Table 12-1 Probability of Observing an Adverse Event

| | | Number of Sul | jects per Treatı | nent Group <sup>b</sup> | |
|---|---|---|---|---|---|
| AE Incidences <sup>a</sup> | 10 | 20 | 30 | 40 | 50 |
| 5% | 40% | 64% | 79% | 87% | 92% |
| 10% | 65% | 88% | 96% | 98% | >99% |
| 15% | 80% | 96% | >99% | >99% | >99% |

AE: adverse event

<sup>a</sup> AE incidences are based on 4 weeks of treatment in Parts 1 and 2,

b Applies to Parts 1

## 12.1.1.2 Efficacy

Table 12-2 provides the power to reject the null within-group hypothesis of no difference in the mean absolute change from baseline for ppFEV<sub>1</sub> through Day 29 or Week 12, as applicable, for any treatment group in Parts 1, 2, with a sample size ranging from 8 to 44 subjects per treatment group. The power calculations are based on a 2-sided 1-sample *t*-test at alpha = 5% using the PASS software package (Version 11.0), assuming an absolute mean change of 3 to 7 percentage points and an SD of 8 percentage points in the absolute change from baseline for ppFEV<sub>1</sub>. Sample sizes of 16 to 44 subjects per treatment group provide adequate power for mean changes of 5 to 7 percentage points as expected in Parts 1, 2,

Table 12-2 Power for Within-group Difference for Mean Absolute Change From Baseline in ppFEV<sub>1</sub>

| Mean Absolute<br>Change From | Number of Subjects per Treatment Group <sup>a</sup> | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Baseline in ppFEV <sub>1</sub> | 8 | 16 | 20 | 22 | 24 | 40 | 42 | 44 |
| 3% | 15% | 29% | 36% | 39% | 42% | 64% | 66% | 68% |
| 4% | 23% | 46% | 56% | 61% | 65% | 87% | 89% | 90% |
| 5% | 33% | 65% | 76% | 80% | 83% | 97% | 98% | 98% |
| 6% | 45% | 80% | 89% | 92% | 94% | >99% | >99% | >99% |
| 7% | 57% | 90% | 96% | 97% | 98% | >99% | >99% | >99% |

ppFEV<sub>1</sub>: forced expiratory volume in 1 second; SD: standard deviation

Note: An SD of 8 percentage points for the absolute change from baseline in ppFEV<sub>1</sub> was used for power calculations.

a Applies to Parts 1

## 12.1.2 Secondary Objectives

A secondary objective of the study is the evaluation of the PD effect of VX-440 in TC with TEZ/IVA (all parts)

# 12.1.2.1 Pharmacodynamic Effect (Part 1)

The absolute change from baseline through Day 29 in sweat chloride is a secondary endpoint used to evaluate the PD objective of the study. In Part 1, a test for a decreasing dose-response trend between placebo and the TC dose groups will be performed using a multiple comparisons procedure (MCP). The procedure consists of testing the null hypothesis of the lack of a decreasing dose-response trend versus a decreasing trend using the 1-sided maximum t-statistic that controls the type I error at alpha = 5%. The procedure requires a family of candidate dose-response models to be prespecified, that covers the range of plausible and diverse dose-response profiles.

The candidate models that best describe the expected decreasing dose-response profile of the TC groups compared to placebo include a linear model, a maximum effect ( $E_{max}$ ) model, and a sigmoid  $E_{max}$  model. The contrasts (i.e., linear combinations of the treatment group means through Day 29) selected to perform the MCP and that capture the shape of these candidate models are described in Table 12-3 below.

Table 12-3 Contrast Coefficients for the Multiple Comparisons Procedure in Part 1, Cohort 1B

| Candidate Model | Placebo | TC-1B-low | TC-1B-high |
|--------------------------|---------|-----------|------------|
| Linear | 1.0 | 0.0 | -1.0 |
| $\mathrm{E}_{max}$ | 1.0 | -0.5 | -0.5 |
| Sigmoid E <sub>max</sub> | 0.5 | 0.5 | -1.0 |

E<sub>max</sub>: maximum effect; TC: triple combination

Table 12-4 provides the power to detect a dose-response trend with the MCP procedure for 3 different expected dose-response profiles with a total sample size of 32 subjects in Cohort 1B assigned to TC-1B-high, TC-1B-low, and placebo in the ratio 2:1:1, based on 5000 simulations for each profile using the MCPMod R software package [Version 1.0-8].

Table 12-4 Power to Detect a Dose-response Trend Based on Change From Baseline in Sweat Chloride in Part 1, Cohort 1B

| Mean Change From Baseline in Sweat Chloride | | | | |
|---|---|---|---|---|
| Candidate Model | Placebo | TC-1B-low | TC-1B-high | Power |
| Linear | 0 | -15 | -20 | 95% |
| Sigmoid E <sub>max</sub> | 0 | 0 | -20 | 99% |
| $\mathrm{E}_{\mathtt{max}}$ | 0 | -20 | -20 | 96% |

E<sub>max</sub>: maximum effect; TC: triple combination

Note: A 1-sided maximum *t*-statistic with a sample size of 32 subjects in Cohort 1B assigned to TC-1B-high, TC-1B-low, and placebo at a ratio 2:1:1 was used for power calculations. An SD change from baseline in sweat chloride of 13 mmol/L was used for power calculations.

Table 12-5 provides the power to reject the null within-group hypothesis of no difference in the mean absolute change from baseline for sweat chloride through Day 29 (Parts 1 and 2) for any treatment group with a sample size ranging from 8 to 44 subjects per treatment group. The power calculations are based on a 2-sided 1-sample *t*-test at alpha = 5% using the PASS software package (Version 11.0), assuming a mean change of -10 to -20 mol/L and an SD of 13 mmol/L in the absolute change from baseline for sweat chloride.

Table 12-5 Power for Within-group Difference for Mean Absolute Change From Baseline in Sweat Chloride

| Mean Absolute Change<br>From Baseline in Sweat | | | Number of | Subjects p | er Treatm | ent Group | 1 | |
|---|---|---|---|---|---|---|---|---|
| Chloride (mmol/L) | 8 | 16 | 20 | 22 | 24 | 40 | 42 | 44 |
| -10 | 47% | 82% | 90% | 93% | 95% | >99% | >99% | >99% |
| -12 | 61% | 93% | 97% | 98% | 99% | >99% | >99% | >99% |
| -15 | 80% | 99% | >99% | >99% | >99% | >99% | >99% | >99% |
| -18 | 92% | >99% | >99% | >99% | >99% | >99% | >99% | >99% |
| -20 | 96% | >99% | >99% | >99% | >99% | >99% | >99% | >99% |

SD: standard deviation

Note: An SD of 13 mmol/L for the absolute change from baseline in sweat chloride was used for power calculations.

Applies to Parts 1

# 12.2 Analysis Sets

The following analysis sets are defined: All Subjects Set, Full Analysis Set, and Safety Set. Additional analysis sets related to the Run-in Period in Part 2 will be defined in the statistical analysis plan, as appropriate.

The **All Subjects Set** will include all subjects who were randomized or received at least 1 dose of study drug. This analysis set will be used for all individual subject data listings and disposition summary tables, unless otherwise specified.

The **Full Analysis Set (FAS)** will include all randomized subjects who have received at least 1 dose of study drug in the Treatment Period. The FAS will be used to summarize subject demographics and baseline characteristics, and for all PD and efficacy analyses, unless otherwise specified.

The **Safety Set** will include all subjects who received at least 1 dose of study drug in the Treatment Period. The Safety Set will be used for all safety analyses, unless otherwise specified.

### 12.3 Statistical Analysis

This section presents a summary of the planned statistical analyses of the primary PD and efficacy endpoints of the study. Statistical analysis details will be provided in the statistical analysis plan (SAP) and clinical pharmacologic analysis details will be provided in the clinical pharmacology analysis plan (CPAP). Both plans will be finalized before the clinical data lock and unblinding of the study.

#### 12.3.1 General Considerations

Continuous variables will be summarized using the following descriptive summary statistics: the number of subjects (n), mean, SD, standard error (SE), median, minimum value (min), and maximum value (max). The precision of the measurement for each continuous variable will be specified in the SAP. Unless otherwise specified, minimum and maximum values will be reported with the same precision as the units of the raw data. The mean, median, SD, and SE will be reported to 1 additional decimal place. Any values that require a transformation to standard units (metric or International System [SI]) will be converted with the appropriate precision.

**Categorical variables** will be summarized using counts and percentages. Percentages will be presented to 1 decimal place.

The **baseline** value, unless otherwise specified, will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the Treatment Period (i.e., Day 1). For ECG, baseline will be defined as the average of the most recent triplicate pretreatment measurements before the first dose of study drug in the Treatment Period (i.e., Day 1).

**Absolute change** from baseline will be calculated as postbaseline value – baseline value.

**Relative change** from baseline will be calculated as (postbaseline value – baseline value)/baseline value.

The Treatment-emergent (TE) Period will include the time from the first dose in the Treatment Period to the Safety Follow-up Visit or 28 days after the last dose of the study drug for subjects who do not complete the Safety Follow-up Visit. Additional TE periods related to the Run-in Period for Part 2 will be defined in the SAP, as appropriate.

There will be no multiplicity adjustment for performing multiple hypothesis tests.

The rules for handling missing data due to treatment or study discontinuation will be described in the SAP.

All data will be summarized for Parts 1, 2, separately, unless specified otherwise.

### 12.3.2 Background Characteristics

# 12.3.2.1 Subject Disposition

The number and percentage of subjects in each disposition category (e.g., randomized, included in the FAS, included in the Safety Set, completed Treatment Period, completed study/Safety Follow-up Visit, and discontinued treatment or study with a breakdown of the reasons for discontinuation) will be summarized overall and by treatment group.

### 12.3.2.2 Demographics and Baseline Characteristics

Demographic, background (e.g., medical history), and baseline characteristics will be summarized using descriptive summary statistics.

The following demographics and baseline characteristics will be summarized overall and by treatment group for the FAS and will include (but are not limited to): sex, race, age, baseline weight, baseline height, baseline BMI, baseline ppFEV<sub>1</sub> and baseline sweat chloride.

No statistical tests will be performed to evaluate baseline imbalance between treatment groups.

#### 12.3.2.3 Prior and Concomitant Medications

Medications used in this study will be coded using the World Health Organization Drug Dictionary Enhanced and categorized as the following:

- **Prior medication:** any medication that started before initial dosing of study drug, regardless of when it ended
- Concomitant medication: medication continued or newly received during the TE Period
- Post-treatment medication: medication continued or newly received after the TE Period

A given medication may be classified as a prior medication, a concomitant medication, or a post-treatment medication; both prior and concomitant; both concomitant and post-treatment; or prior, concomitant, and post-treatment. If a medication has a missing or partially missing start/end date or time and if it cannot be determined whether it was taken before the first dose of study drug, concomitantly during the TE Period, or after the TE Period, it will be considered in all 3 categories of prior, concomitant, and post-treatment medication.

Prior medications and concomitant medications will be summarized descriptively by Preferred Name based on the FAS. Post-treatment medications will be provided separately in an individual subject data listing.

Additional classifications of concomitant medications related to the Run-in Period will be defined in the SAP, as appropriate.

# 12.3.2.4 Study Drug Exposure and Compliance

Exposure to study drug will be summarized for the FAS in terms of duration of treatment a subject received (in days), defined as the last day minus the first day of study drug plus 1.

Dosing compliance based on number of pills taken, will be summarized for the FAS, and will be derived as  $100 \times [(\text{total number of pills dispensed}) - (\text{total number of pills returned})]/(\text{total number of pills planned to be taken per day} \times \text{duration of study drug exposure in days}).$ 

Dosing compliance based on study drug exposure, will be derived as  $100 \times [1 - (total number of days of study drug interruption) / (duration of study drug exposure in days)].$ 

### 12.3.2.5 Important Protocol Deviations

An important protocol deviation (IPD) is a deviation that may significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. The rules for identifying an IPD will be described in the SAP.

All IPDs will be provided in an individual subject data listing.

A coprimary objective of the study is the evaluation of the efficacy of

## 12.3.3 Efficacy Analysis

VX-440 in TC with TEZ/IVA (all parts). 12.3.3.1 **Analysis of Primary Efficacy Variables** The primary efficacy variable is the absolute change from baseline for ppFEV<sub>1</sub> through Day 29 The analysis will be performed using a mixedin Parts 1 and 2, effects model for repeated measures (MMRM) with change from baseline as the dependent variable. stratification factors at randomization as categorical covariates, when applicable. The model will be estimated using restricted maximum likelihood. Denominator degrees of freedom for the F test for fixed effects will be estimated using the Kenward-Roger approximation. A compound symmetry covariance structure will be used to model the within-subject errors. Conditional on fixed effects, missing data due to treatment or study discontinuation will be assumed to be missing at random. Descriptive analyses of the change from baseline will be performed for all treatment groups in Adjusted means and 95% confidence intervals of the average treatment effects through Day 29 or Week 12, as applicable, with 2-sided P values, will be estimated within MMRM using LSMeans via PROC MIXED in SAS, for all within-group and between-group comparisons in all parts. Further, relevant data from Parts 1, 2, will be pooled as appropriate within MMRM with appropriate adjustment for covariates. Details will be provided in the SAP.

There will be no multiplicity adjustment for performing multiple hypothesis tests.

# 12.3.3.2 Analysis of Secondary Efficacy Variables

The secondary efficacy variables include:

| • | Relative change in ppFEV <sub>1</sub> from baseline through Day 29 (Parts 1 and 2) and |
|---|---|
| • | Absolute change in the CFQ-R respiratory domain score from baseline at Day 29 (Parts 1 and 2) |

Details of the analysis will be provided in the SAP.



## 12.3.4 Pharmacodynamic Analysis

A secondary objective of the study is the evaluation of the PD effect on sweat chloride concentrations of VX-440 in TC with TEZ/IVA (all parts).

# 12.3.4.1 Pharmacodynamic Effect

The absolute change in sweat chloride from baseline through Day 29 is a secondary endpoint used to evaluate the PD objective of the study. The test to detect a decreasing dose-response trend of VX-440 at 2 doses in TC with TEZ/IVA relative to placebo based on sweat chloride, will be performed using the MCP procedure with the prespecified comparisons (contrasts) of the treatment group means within a linear MMRM framework. The model will include treatment group, visit, and treatment-by-visit interaction as fixed effects, with the ppFEV<sub>1</sub> stratification factor at randomization as a categorical covariate. The test will be performed using the 1-sided maximum t-statistic of the individual t-statistics for the multiple prespecified contrasts at alpha = 5%, based on the treatment group means through Day 29 in Cohort 1B.



Adjusted means and 95% confidence intervals of the average treatment effects through Day 29 or Week 12, as applicable, with 2-sided *P* values, for all within-group and between-group

comparisons in all parts will be estimated within MMRM, with appropriate adjustment for covariates.

Additional details of the analysis will be provided in the SAP.

### 12.3.5 Safety Analysis

A coprimary objective of the study is the evaluation of safety and tolerability. All safety analyses will be based on data from the TE Period for all subjects in the Safety Set.

The overall safety profile of study drug will be assessed based on the following safety and tolerability endpoints:

- Treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (i.e., hematology, serum chemistry, coagulation, and urinalysis)
- ECGs
- Vital signs
- Pulse oximetry

All safety data will be summarized by treatment group and overall, for each Part.

All safety data will be presented in individual subject data listings.

#### 12.3.5.1 Adverse Events

For analysis purposes, AEs will be classified as pretreatment AEs, TEAEs, or post-treatment AEs, defined as follows:

- Pretreatment AE: any AE that started before the first dose of study drug
- TEAE: any AE that increased in severity or that was newly developed at or after the first dose of study drug through the end of the TE Period
- Post-treatment AE: any AE that increased in severity or that was newly developed beyond the TE Period

For AEs with missing or partial start dates, if there is no clear evidence that the AEs started before or after study drug treatment, then the AEs will be classified as TEAEs.

AE summary tables will be presented for TEAEs only, overall and by treatment group for each Part, and will include the following:

- All TEAEs
- TEAEs by strongest relationship
- TEAEs by maximum severity
- TEAEs leading to treatment discontinuation
- Serious TEAEs
- TEAEs leading to death
- Frequently reported TEAEs

Summaries will be presented by MedDRA system organ class and preferred term using frequency counts and percentages (i.e., number and percentage of subjects with an event). When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, only the maximum severity level will be presented in the severity summaries, and the strongest relationship level in the relationship summaries. In addition, a listing containing individual subject level AE data for all deaths and other serious and significant AEs will be provided separately. All AEs, including pre- and post-treatment AEs, will be presented in individual subject data listings.

### 12.3.5.2 Clinical Laboratory Assessments

For the treatment-emergent laboratory measurements, the observed values and change from baseline values of the continuous hematology, chemistry, and coagulation results will be summarized in SI units overall and by treatment group at each scheduled visit.

The number and percentage of subjects meeting a threshold analysis criterion during the TE Period will be summarized overall and by treatment group for each part. The threshold analysis criterion shift from baseline will also be summarized for selected laboratory parameters. The threshold analysis criteria and the parameter selection criteria will be provided in the SAP.

Results of urinalysis and the serum pregnancy test will be listed in individual subject data listings only. In addition, a listing containing individual subject hematology, chemistry, and coagulation values outside the reference ranges will be provided. This listing will include data from scheduled and unscheduled visits.

# 12.3.5.3 Electrocardiogram

For the treatment-emergent ECG measurements, a summary of observed values and change from baseline values will be provided overall and by treatment group for each Part, at each scheduled visit and time point, as applicable, for the following ECG interval measurements (in ms): RR, PR, QT, and QT corrected for HR (QTcF), QRS duration, and HR (beats per minute).

The number and percentage of subjects meeting a threshold analysis criterion during the TE Period will be summarized overall and by treatment group. The threshold analysis criteria will be provided in the SAP.

Additional ECG analyses will be described in the SAP.

#### 12.3.5.4 Vital Signs

For the treatment-emergent vital signs measurements, the observed values and change from baseline values will be summarized overall and by treatment group at each scheduled visit. The following vital signs parameters will be summarized: systolic and diastolic blood pressure (mm Hg), body temperature (°C), HR (beats per minute), and respiratory rate (breaths per minute).

The number and percentage of subjects meeting a threshold analysis criterion during the TE Period will be summarized overall and by treatment group for each part. The threshold analysis criteria will be provided in the SAP.

Additional vital signs analyses will be described in the SAP.

# 12.3.5.5 Pulse Oximetry

For the treatment-emergent pulse oximetry measurements, a summary of observed values and change from baseline values will be provided overall and by treatment group for each Part, at each scheduled visit for the percent of oxygen saturation by pulse oximetry.

The number and percentage of subjects with shift changes from baseline (normal/missing and low according to the reference range) to the lowest percent of oxygen saturation during the TE Period will be summarized overall and by treatment group.

## 12.3.5.6 Physical Examination

PE findings will be presented in an individual subject data listing only.

### 12.3.5.7 Other Safety Analysis

Not applicable.

### 12.3.6 Interim and IDMC Analyses

## 12.3.6.1 Interim Analysis

Separate interim analyses will be performed after:

- all subjects in Part 1 have completed the Safety Follow-up Visit
- all subjects in Part 2 have completed the Safety Follow-up Visit

The interim results of Parts 1 and 2 will be unblinded for full review by the Vertex study team.

## 12.3.6.2 IDMC Analysis

The safety of the TC will be monitored by an external, IDMC to ensure the safety of the subjects in the study.

An IDMC will be formed before study initiation. The IDMC's objectives, responsibilities, and operational details will be defined in a separate document (IDMC Charter), which will be finalized before the first subject is randomized in the study. The IDMC will conduct planned safety reviews of study data from all parts of the study as outlined in the IDMC Charter.

## 12.4 Clinical Pharmacology Analysis

## 12.4.1 Pharmacokinetic Analysis

The PK analysis of VX-440, TEZ and metabolite M1-TEZ, and IVA and metabolite M1-IVA will be performed using nonlinear mixed effects modeling. Standard noncompartmental analysis may also be performed as data allow. Descriptive statistics will be used to summarize PK parameter values for all analytes.

A detailed description of the planned PK analysis will be presented in the CPAP.

# 12.4.2 Pharmacokinetic/Pharmacodynamic Analyses

PD assessments to be included in PK/PD analyses may include sweat chloride, ppFEV<sub>1</sub>, as well as other secondary endpoints such as CFQ-R. Comparison between postdose and predose values will be performed and expressed as a change from baseline.

A sequential approach will be used to perform the population PK/PD analysis. The Bayesian estimates of individual PK parameters from the final population PK model will be used to
simulate PK profiles for each subject. The simulated VX-440, TEZ, IVA, or metabolite plasma concentrations will be used in the potential pharmacological response models to describe changes in each endpoint from baseline. Fixed- and random-effect parameter estimates and the associated asymptotic SEs will be estimated. Descriptive statistics will be used to summarize Bayesian estimates of individual PK/PD parameters obtained from the population PK/PD model.

## 13 PROCEDURAL, ETHICAL, REGULATORY, AND ADMINISTRATIVE CONSIDERATIONS

# 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting

#### 13.1.1 Adverse Events

#### 13.1.1.1 Definition of an Adverse Event

An AE is defined as any untoward medical occurrence in a subject during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or worsening of a pre-existing condition (e.g., increase in its severity or frequency) after the ICF is signed.

An AE is considered serious if it meets the definition in Section 13.1.2.1.

### 13.1.1.2 Clinically Significant Assessments

Study assessments including laboratory tests, ECGs, PEs, and vital signs will be assessed and those deemed to have clinically-significant worsening from baseline will be documented as an AE. When possible, a clinical diagnosis for the study assessment will be provided, rather than the abnormal test result alone (e.g., urinary tract infection, anemia). In the absence of a diagnosis, the abnormal study assessment itself will be listed as the AE (e.g., bacteria in urine or decreased hemoglobin).

An abnormal study assessment is considered clinically significant if the subject has 1 or more of the following:

- Concomitant signs or symptoms related to the abnormal study assessment
- Further diagnostic testing or medical/surgical intervention
- A change in the dose of study drug or discontinuation from the study

Repeat testing to determine whether the result is abnormal, in the absence of any of the above criteria, does not necessarily meet clinically significant criteria. The determination of whether the study assessment results are clinically significant will be made by the investigator.

A laboratory value that is Grade 4 will not automatically be an SAE. A Grade 4 laboratory value will be an SAE if the subject's clinical status indicates a life-threatening AE.

#### 13.1.1.3 Documentation of Adverse Events

All AEs will be collected from the time ICF is signed until the following time points:

 For subjects who do not enroll: until time of screen failure (e.g., screen failure, withdrawal of consent)

- For enrolled subjects who have a Safety Follow-up Visit: through the Safety Follow-up Visit
- For enrolled subjects who do not have a Safety Follow-up Visit, the earliest of
  - o 28 days after the last dose of study drug, or
  - o the ETT Visit, if that visit is 3 weeks or later following the last dose of study drug (see Section 8.1.6).

All subjects will be queried, using nonleading questions, about the occurrence of AEs at each study visit. When possible, a constellation of signs and/or symptoms will be identified as 1 overall event or diagnosis. All AEs for enrolled subjects will be recorded in the CRF and source document. AEs for subjects who are screened but not subsequently enrolled in the study will be recorded only in the subject's source documents. The following data will be documented for each AE:

- Description of the event
- Classification of "serious" or "nonserious"
- Date of first occurrence and date of resolution (if applicable)
- Severity
- Causal relationship to study drug(s)
- Action taken
- Outcome
- Concomitant medication or other treatment given

#### 13.1.1.4 Adverse Event Severity

The investigator will determine and record the severity of all serious and nonserious AEs. The guidance available at the following website will be consulted: Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03, Cancer Therapy Evaluation Program, http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm (Accessed August 2015). AEs of CTCAE Grades 4 and 5 will be documented as "life-threatening." In considering the severity of an AE in a pediatric subject, the investigator will consider that reference ranges for pediatric clinical laboratory parameters may differ from those given in the CTCAE. The severity of an AE that does not appear in the CTCAE will be determined according to the definitions in Table 13-1.

Table 13-1 Grading of AE Severity

| Classification | Definition |
|---|---|
| Mild (Grade 1) | Mild level of discomfort and does not interfere with regular activities |
| Moderate (Grade 2) | Moderate level of discomfort and significantly interferes with regular activities |
| Severe (Grade 3) | Significant level of discomfort and prevents regular activities |
| Life-threatening (Grade 4) | Any adverse drug event that places the subject, in the view of the investigator, at immediate risk of death |

## 13.1.1.5 Adverse Event Causality

Every effort will be made by the investigator to assess the relationship of the AE, if any, to the study drug(s). Causality will be classified using the categories presented in Table 13-2.

Table 13-2 Classifications for AE Causality

| Classification | Definition |
|---|---|
| Related | There is an association between the event and the administration of investigational study drug, a plausible mechanism for the event to be related to the investigational study drug and causes other than the investigational study drug have been ruled out, and/or the event reappeared on re-exposure to the investigational study drug. |
| Possibly related | There is an association between the event and the administration of the investigational study drug and there is a plausible mechanism for the event to be related to investigational study drug, but there may also be alternative etiology, such as characteristics of the subject's clinical status or underlying disease. |
| Unlikely related | The event is unlikely to be related to the investigational study drug and likely to be related to factors other than investigational study drug. |
| Not related | The event is related to an etiology other than the investigational study drug (the alternative etiology will be documented in the study subject's medical record). |

## 13.1.1.6 Study Drug Action Taken

The investigator will classify the study drug action taken with regard to the AE. The action taken will be classified according to the categories shown in Table 13-3.

Table 13-3 Classifications for Study Drug Action Taken With Regard to an AE

| Classification | Definition |
|---|---|
| Dose not changed | Study drug dose not changed in response to an AE |
| Dose reduced | Study drug dose reduced in response to an AE |
| Drug interrupted Study drug administration interrupted in response to an AE | |
| <b>Drug withdrawn</b> Study drug administration permanently discontinued in response to an AE | |
| Not applicable | Action taken regarding study drug administration does not apply. |
| | "Not applicable" will be used in circumstances such as when the investigational treatment had been completed before the AE began and no opportunity to decide whether to continue, interrupt, or withdraw treatment is possible. |

AE: adverse event

#### 13.1.1.7 Adverse Event Outcome

An AE will be followed until the investigator has determined and provided the final outcome. The outcome will be classified according to the categories shown in Table 13-4.

Table 13-4 Classifications for Outcome of an AE

| Classification | Definition |
|---|---|
| Recovered/Resolved | Resolution of an AE with no residual signs or symptoms |
| Recovered/Resolved With Sequelae | Resolution of an AE with residual signs or symptoms |
| Not Recovered/Not<br>Resolved (Continuing) | Either incomplete improvement or no improvement of an AE, such that it remains ongoing |

Vertex Pharmaceuticals Incorporated

Table 13-4 Classifications for Outcome of an AE

| Classification | Definition |
|---|---|
| Fatal | Outcome of an AE is death. "Fatal" will be used when death is at least possibly related to the AE. |
| Unknown | Outcome of an AE is not known (e.g., a subject lost to follow-up) |

AE: adverse event

#### 13.1.1.8 Treatment Given

The investigator ensures adequate medical care is provided to subjects for any AEs, including clinically significant laboratory values related to study drug. In addition, the investigator will describe whether any treatment was given for the AE. "Yes" is used if any treatment was given in response to an AE, and may include treatments such as other medications, hospitalization, surgery, or physical therapy. "No" indicates the absence of any kind of treatment for an AE.

#### 13.1.2 Serious Adverse Events

#### 13.1.2.1 Definition of a Serious Adverse Event

An SAE is any AE that meets any of the following outcomes:

- Fatal (death, regardless of cause, that occurs during participation in the study or occurs after
  participation in the study and is suspected of being a delayed toxicity due to administration of
  the study drug)
- Life-threatening, such that the subject was at immediate risk of death from the reaction as it occurred
- Inpatient hospitalization or prolongation of hospitalization
- Persistent or significant disability/incapacity (disability is defined as a substantial disruption of a person's ability to conduct normal life functions)
- Congenital anomaly or birth defect
- Important medical event that, based upon appropriate medical judgment, may jeopardize the subject or may require medical or surgical intervention to prevent 1 of the outcomes listed above (e.g., an allergic bronchospasm requiring intensive treatment in an emergency room or at home)

If a subject has a hospitalization or procedure (e.g., surgery) for an event or condition that occurred before the subject signed the ICF, and the hospitalization or procedure was planned before the subject signed the ICF, the hospitalization or procedure will not be considered to indicate an SAE, unless an AE caused the hospitalization or procedure to be rescheduled sooner or to be prolonged relative to what was planned. In addition, hospitalizations clearly not associated with an AE (e.g., social hospitalization for purposes of respite care) will not be considered to indicate an SAE.

Clarification will be made between the terms "serious" and "severe" because they are not synonymous. The term "severe" is often used to describe the intensity (severity) of a specific event, as in mild, moderate, or severe myocardial infarction. The event itself, however, may be of relatively minor medical significance, such as a severe headache. This is not the same as

"serious," which is based on subject/event outcome or action described above, and is usually associated with events that pose a threat to a subject's life or functioning. Seriousness, not severity, serves as a guide for defining expedited regulatory reporting obligations.

#### 13.1.2.2 Documentation of Serious Adverse Events

All SAEs that occur after obtaining informed consent and assent (where applicable) through the Safety Follow-up Visit, regardless of causality, will be reported by the investigator to Vertex GPS. In addition, all SAEs that occur after the Safety Follow-up Visit and are considered related to study drug(s) will be reported to Vertex GPS within 24 hours.

SAEs will be recorded on the Vertex Organized Safety Information Collection Form (hereafter referred to as the "SAE Form") using a recognized medical term or diagnosis that accurately reflects the event. SAEs will be assessed by the investigator for relationship to the investigational study drug(s) and possible etiologies. On the SAE Form, relationship to study drug(s) will be assessed only as related (includes possibly related) or not related (includes unlikely related), and severity assessment will not be required. For the purposes of study analysis, if the event has not resolved at the end of the study reporting period, it will be documented as ongoing. For purposes of regulatory safety monitoring, the investigator is required to follow the event to resolution and report to Vertex the outcome of the event using the SAE Form.

#### 13.1.2.3 Reporting Serious Adverse Events

The investigator is responsible for notifying the sponsor within 24 hours of identifying an SAE, regardless of the presumed relationship to the investigational study drug. The SAE Form will be completed for new/initial events as well as to report follow-up information on previously reported events. Investigators are asked to report follow-up information as soon as it becomes available to ensure timely reporting to health authorities.

Please send completed SAE Forms to Vertex GPS via:

| Email: | (preferred choice) |
|--------------------|--------------------|
| Fax: | |
| Contact Telephone: | |

## 13.1.2.4 Expedited Reporting and Investigator Safety Letters

Vertex, as study sponsor, is responsible for reporting suspected, unexpected, serious adverse reactions (SUSARs) involving the study drug(s) to all regulatory authorities and participating investigators in accordance with ICH Guidelines and/or local regulatory requirements, as applicable. In addition, Vertex, or authorized designee, will be responsible for the submission of safety letters to central independent ethics committees (IECs).

It is the responsibility of the investigator or designee to promptly notify the local institutional review board (IRB)/local IEC of all unexpected serious adverse drug reactions involving risk to human subjects.

## 13.2 Administrative Requirements

#### 13.2.1 Ethical Considerations

The study will be conducted in accordance with the current ICH GCP Guidelines, which are consistent with the ethical principles founded in the Declaration of Helsinki, and in accordance

with local applicable laws and regulations. The IRB/IEC will review all appropriate study documentation to safeguard the rights, safety, and well-being of the subjects. The study will only be conducted at sites where IRB/IEC approval has been obtained. The protocol, Investigator's Brochure, sample ICF, advertisements (if applicable), written information given to the subjects (including diary cards), safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB/IEC by the investigator or Vertex, as allowable by local applicable laws and regulations.

### 13.2.2 Subject Information and Informed Consent

After the study has been fully explained, written informed consent will be obtained from the subject or legal representative or guardian (if applicable), and assent will be obtained from the subject (if applicable), before study participation. The method of obtaining and documenting the informed consent and assent (if applicable) and the contents of the consent will comply with ICH GCP and all applicable laws and regulations and will be subject to approval by Vertex or its designee.

## 13.2.3 Investigator Compliance

No modifications to the protocol will be made without the approval of both the investigator and Vertex. Changes that significantly affect the safety of the subjects, the scope of the investigation, or the scientific quality of the study (i.e., efficacy assessments) will require IRB/IEC notification before implementation, except where the modification is necessary to eliminate an apparent immediate hazard to human subjects. Vertex will submit all protocol modifications to the required regulatory authorities.

When circumstances require an immediate departure from procedures set forth in the protocol, the investigator will contact Vertex to discuss the planned course of action. If possible, contact will be made before the implementation of any changes. Any departures from the protocol will be fully documented in the source documentation and in a protocol deviation log.

#### 13.2.4 Access to Records

The investigator will make the office and/or hospital records of subjects enrolled in this study available for inspection by Vertex or its representative at the time of each monitoring visit and for audits. The records will also be available for direct inspection, verification, and copying, as required by applicable laws and regulations, by officials of the regulatory health authorities (FDA and others). The investigator will comply with applicable privacy and security laws for use and disclosure of information related to the research set forth in this protocol.

### 13.2.5 Subject Privacy

To maintain subject confidentiality and to comply with applicable data protection and privacy laws and regulations, all CRFs, study reports, and communications relating to the study will identify subjects by assigned subject numbers and access to subject names linked to such numbers shall be limited to the site and the study physician and shall not be disclosed to Vertex. As required by applicable laws and regulations in the countries in which the study is being conducted, the investigator will allow Vertex and/or its representatives access to all pertinent medical records to allow for the verification of data gathered in the CRFs/SAE forms and the review of the data collection process. The FDA and regulatory authorities in other jurisdictions, including the IRB/IEC, may also request access to all study records, including source documentation, for inspection.

For sites participating in the study in the US, and in accordance with the Health Insurance Portability and Accountability Act and associated regulations ("HIPAA") an executed HIPAA authorization shall be obtained by the site from each subject (or the legal representative of the subject) before research activities may begin. Each HIPAA authorization shall comply with all HIPAA requirements including authorization allowing the site access to and use of the subject's personally identifiable health information, authorization for the site to disclose such information to Vertex, the FDA, and other parties requiring access under the protocol, and statements as to the purpose for which such information may be used and for how long.

#### 13.2.6 Record Retention

The investigator will maintain all study records according to ICH GCP guidelines and/or applicable local regulatory requirement(s), whichever is longest, as described in the Clinical Trial Agreement. If the investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility and Vertex will be notified.

#### 13.2.7 Study Termination

At any time, Vertex may terminate this study in its entirety or may terminate this study at any particular site. In addition, for reasonable cause, either the investigators or their IRBs/IECs may terminate the study at their center.

Conditions that may lead to reasonable cause and warrant termination include, but are not limited to:

- Subject or investigator noncompliance
- Unsatisfactory subject enrollment
- Lack of adherence to protocol procedures
- Lack of evaluable and/or complete data
- Potentially unacceptable risk to study subjects
- Decision to modify drug development plan
- Decision by the FDA or other regulatory authority

Written notification that includes the reason for the clinical study termination is required.

## 13.3 Data Quality Assurance

Vertex or its designated representative will conduct a study site visit to verify the qualifications of each investigator, inspect clinical study site facilities, and inform the investigator of responsibilities and procedures for ensuring adequate and correct study documentation.

The investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each study participant. Study data for each enrolled subject will be entered into a CRF by study site personnel using a secure, validated, web-based electronic data capture (EDC) application. Vertex will have read-only access to site-entered clinical data in the EDC application.

Instances of missing, discrepant, or uninterpretable data will be queried with the investigator for resolution. Any changes to study data will be made to the CRF and documented in an audit trail, which will be maintained within the clinical database.

## 13.4 Monitoring

Monitoring and auditing procedures developed or approved by Vertex will be followed to comply with GCP guidelines. On-site checking of the CRFs/SAE Forms for completeness and clarity, cross-checking with source documents, and clarification of administrative matters will be performed.

The study will be monitored by Vertex or its designee. Monitoring will be done by personal visits from a representative of Vertex, or designee (study site monitor), who will review the CRFs/SAE Forms and source documents. The study site monitor will ensure that the investigation is conducted according to the protocol design and regulatory requirements.

## 13.5 Electronic Data Capture

Vertex will provide the study sites with secure access to and training on the EDC application sufficient to permit study site personnel to enter or correct information in the CRFs on the subjects for which they are responsible.

A CRF will be completed for each enrolled study subject. It is the investigator's responsibility to ensure the accuracy, completeness, clarity, and timeliness of the data reported in the subject's CRF. Source documentation supporting the CRF data will indicate the subject's participation in the study and will document the dates and details of study procedures, AEs, other observations, and subject status.

The investigator, or designated representative, will complete the CRF as soon as possible after information is collected.

The audit trail entry will show the user's identification information and the date and time of any correction. The investigator will provide formal approval of all the information in the CRFs, including any changes made to the CRFs, to endorse the final submitted data for the subjects for whom the investigator is responsible.

Vertex will retain the CRF data and corresponding audit trails. A copy of the final archival CRF in the form of a CD or other electronic media will be placed in the investigator's study file.

## 13.6 Publications and Clinical Study Report





## 13.6.2 Clinical Study Report

A clinical study report, written in accordance with the ICH E3 Guideline, will be submitted in accordance with local regulations.

#### 14 REFERENCES

- 1 Cystic Fibrosis Foundation. About CF. Available at: http://www.cff.org/AboutCF/. Accessed 30 June 2015.
- 2 Kreindler JL. Cystic fibrosis: exploiting its genetic basis in the hunt for new therapies. Pharmacol Ther. 2010;125(2):219-29.
- Development FOoOP. Developing Products for Rare Diseases & Conditions [Internet]. Available from: http://www.fda.gov/ForIndustry/DevelopingProductsforRareDiseasesConditions/default. htm. . Accessed
- Agency EM. Committee for Orphan Medicinal Products (COMP) [Internet]. Available from:

  http://www.ema.europa.eu/ema/index.jsp?curl=pages/about\_us/general/general\_content\_
  000263.jsp&murl=menus/about\_us/about\_us.jsp&mid=WC0b01ac0580028e30.
  Accessed
- 5 Sheppard MN, Nicholson AG. The pathology of cystic fibrosis. Curr Diagn Pathol. 2002;8(1):50-9.
- 6 Cystic Fibrosis Foundation. Patient Registry: 2014 Annual Data Report. Bethesda, MD: Cystic Fibrosis Foundation; 2015.
- Vertex Pharmaceuticals Incorporated. Ivacaftor (VX-770) Investigator's Brochure, Version 12.0. Report date: 08 May 2015.
- 8 Vertex Pharmaceuticals Incorporated. VX-440 Investigator's Brochure, Version 1.0. Report date: 30 September 2015.
- Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, et al. Standardisation of spirometry. Eur Respir J. 2005;26(2):319-38.
- 11 Vertex Pharmaceuticals Incorporated. VX-661 Investigator's Brochure, Version 7.0. Report date: 08 May 2015.
- 12 Vertex Pharmaceuticals Incorporated. Ivacaftor Investigator's Brochure, Version 12.0. Report date: 8 May 2015.
- Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.
- Levey AS, Bosch JP, Lewis JB, Green T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Ann Intern Med. 1999;130(6):461-70.
- Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006;145(4):247-54.
- 16 Counahan R, Chantler C, Ghazali S, Kirkwood B, Rose F, Barratt T. Estimation of glomerular filtration rate from plasma creatinine concentration in children. Arch Dis Child. 1976;51(11):875-8.

- 17 Quittner AL, Buu A, Messer MA, Modi AC, Watrous M. Development and validation of the Cystic Fibrosis Questionnaire in the United States: a health-related quality-of-life measure for cystic fibrosis. Chest. 2005;128(4):2347-54.
- Goss CH, Quittner AL. Patient-reported outcomes in cystic fibrosis. Proc Am Thorac Soc. 2007;4(4):378-86.
- Wenninger K, Aussage P, Wahn U, Staab D. German Cystic Fibrosis Questionnaire study group. The revised German Cystic Fibrosis Questionnaire: validation of a diseasespecific health-related quality of life instrument. Qual Life Res. 2003;12(1):77-85.
- Henry B, Aussage P, Grosskopf C, Goehrs JM. Development of the Cystic Fibrosis Questionnaire (CFQ) for assessing quality of life in pediatric and adult patients. Qual Life Res. 2003;12(1):63-76.
- 21 Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Dřevínek P, et al. A CFTR potentiator in patients with cystic fibrosis and the *G551D* mutation. N Engl J Med. 2011;365(18):1663-72.
- Fuchs HJ, Borowitz DS, Christiansen DH, Morris EM, Nash ML, Ramsey BW, et al. Effect of aerosolized recombinant human DNase on exacerbations of respiratory symptoms and on pulmonary function in patients with cystic fibrosis. N Engl J Med.
- Heads of Medicines Agencies CTFG. Recommendations related to contraception and pregnancy testing in clinical trials. [Internet]. Available from: Accessed 15 September 2014.

## APPENDIX A CFTR Mutations That Are Predicted to Result in a CFTR Protein With Minimal Function (Part 1

Per the study eligibility criteria, heterozygous *F508del-CFTR* subjects in Parts 1 must have a second *CFTR* allele containing a mutation that is predicted to result in a CFTR protein with minimal function and not likely to respond to TEZ and/or ivacaftor (IVA) therapy. These *CFTR* mutations were defined using 3 major sources:

- biological plausibility for the mutation to respond (i.e., mutation class)
- evidence of clinical severity on a population basis (per CFTR2 patient registry; accessed on 15 February 2016)
  - o average sweat chloride >86 mmol/L, and
  - o prevalence of pancreatic insufficiency (PI) >50%
- in vitro testing
  - mutations resulting in baseline chloride transport <10% of wild-type CFTR were considered minimal function
  - o mutations resulting in chloride transport <10% of wild-type CFTR following the addition of TEZ and/or IVA were considered nonresponsive

The clinical severity criteria (average sweat chloride >86 mmol/L and %PI >50%) do not apply to the individual subjects to be enrolled in this study, but were used to classify the mutation status on a population level.

The list below represents acceptable mutations, which are detectable by an FDA-cleared genotyping assay; however, this list may not include every eligible mutation, and investigators should contact the medical monitor regarding other mutations that may also meet study eligibility criteria.

CFTR Mutations Eligible for VX15-440-101, Parts 1

| Criteria | Mutation | | | | |
|---|---|---|---|---|---|
| Truncation mutations | S4X | C276X | G542X | R792X | E1104X |
| <ul> <li>%PI &gt;50% and/or</li> </ul> | G27X | Q290X | | | R1158X |
| SwCl <sup>-</sup> >86 mmol/L | Q39X | G330X | Q552X | W846X | R1162X |
| <ul> <li>no full-length protein</li> </ul> | W57X | W401X | R553X | Y849X | S1196X |
| | E60X | Q414X | E585X | R851X | W1204X |
| | R75X | S434X | G673X | Q890X | L1254X |
| | E92X | S466X | Q685X | S912X | S1255X |
| | Q98X | S489X | R709X | Y913X | W1282X |
| | Y122X | Q493X | K710X | W1089X | Q1313X |
| | E193X | W496X | L732X | Y1092X | E1371X |
| | L218X | C524X | R764X | W1098X | Q1382X |
| | Q220X | Q525X | R785X | R1102X | Q1411X |
| Splice mutations | 185+1G→T | 711+5G→A | A 1717-8G→A | 2622+1G→A | 3121-1G→A |
| <ul> <li>%PI &gt;50% and/or</li> </ul> | 296+1G→A | 712-1G→T | 1717-1G→A | 2790-1G→C | 3500-2A→G |
| SwCl <sup>-</sup> >86 mmol/L | 405+1G→A | 1248+1G→ | A 1811+1G→C | 3040G→C | 3600+2insT |
| no or little mature | 405+3A→C | 1249-1G→ | A 1811+1.6kbA→G | (G970R) | 3850-1G→A |
| mRNA | 406 <b>-</b> 1G→A | 1341+1G→ | A 1812-1G→A | 3120G→A | 4005+1G→A |
| | 621+1G→T | 1525-2A→ | G 1898+1G→A | 3120+1G→A | 4374+1G→T |
| | 711+1G→T | 1525-1G→ | A 1898+1G→C | 3121-2A→G | |
| Small (≤3 nucleotide) | 182delT | 1119delA | 1782delA | 2732insA | 3876delA |
| insertion/deletion (ins/del) | 306insA | 1138insG | 1824delA | 2869insG | 3878delG |
| frameshift mutations | 365-366insT | 1154insTC | 2043delG | 2896insAG | 3905insT |
| • %PI >50% and/or<br>SwCl >86 mmol/L | 394delTT | 1161delC | 2143delT | 2942insT | 4016insT |
| • garbled and/or | 442delA | 1213delT | $2183AA \rightarrow G^a$ | 2957delT | 4021dupT |
| truncated protein | 444delA | 1259insA | 2184delA | 3007delG | 4040delA |
| araneatea protein | 457TAT→G | 1288insTA | 2184insA | 3028delA | 4279insA |
| | 541delC | 1471delA | 2307insA | 3171delC | 4326delTC |
| | 574delA | 1497delGG | 2347delG | 3659delC | |
| | 663delT | 1548delG | 2585delT | 3737delA | |
| | 935delA | 1609del CA | 2594delGT | 3791delC | |
| | 1078delT | 1677delTA | 2711delT | 3821delT | |
| Non-small (>3 nucleotide) | CFTRdele2,3 | 1 | 1461ins4 | 2991del32 | |
| insertion/deletion (ins/del) | CFTRdele22,2 | 23 | 1924del7 | 3667ins4 | |
| frameshift mutations | 124del23bp | 2 | 2055del9→A | 4010del4 | |
| • %PI >50% and/or | 852del22 | | 2105- | 4209TGTT→AA | |
| SwCl >86 mmol/L | | 2 | 2117del13insAGAAA | | |
| <ul> <li>garbled and/or truncated protein</li> </ul> | 991del5 27 | | 2721del11 | | |

## CFTR Mutations Eligible for VX15-440-101, Parts 1

| Criteria | Mutation | | | |
|---|---|---|---|---|
| Class II, III, IV mutations not responsive to IVA alone or in combination with TEZ or LUM • %PI>50% and/or SwCI >86 mmol/L AND • Not responsive in vitro to IVA alone or in combination with TEZ or LUM | A46D <sup>b</sup><br>G85E<br>R347P<br>L467P <sup>b</sup><br>I507del | V520F<br>A559T <sup>b</sup><br>R560T<br>R560S<br>A561E | Y569D <sup>b</sup><br>L1065P<br>R1066C<br>L1077P <sup>b</sup><br>M1101K | N1303K |

CFTR: cystic fibrosis transmembrane conductance regulator; IVA: ivacaftor; LUM: lumacaftor; PI: pancreatic insufficiency; SwCl<sup>-</sup>: sweat chloride; TEZ: tezacaftor

Source: CFTR2.org [Internet]. Baltimore (MD): Clinical and functional translation of CFTR. The Clinical and Functional Translation of CFTR (CFTR2), US Cystic Fibrosis Foundation, Johns Hopkins University, the Hospital for Sick Children. Available at: http://www.cftr2.org/. Accessed 15 February 2016.

<sup>%</sup>PI: percentage of *F508del-CFTR* heterozygous patients in the CFTR2 patient registry who are pancreatic insufficient; SwCI: mean sweat chloride of *F508del-CFTR* heterozygous patients in the CFTR2 patient registry

<sup>&</sup>lt;sup>a</sup> Also known as 2183delAA→G.

b Unpublished data.

## 15 PROTOCOL SIGNATURE PAGES

## 15.1 Sponsor Signature Page

| Protocol #: VX15-440-101 | Version #: | 2.0 | Version Date: | 16 September 2016 |
|---|---|---|---|---|
| Study Title: A Phase 2, Randomiz<br>and Efficacy of VX-440 Combina<br>Cystic Fibrosis | , | - | • | • |

This Clinical Study Protocol has been reviewed and approved by the sponsor.



## 15.2 Investigator Signature Page

| Protocol #: VX15-440-101 | Version #: | 2.0 | Version Date: | 16 September 2016 |
|---|---|---|---|---|
| Study Title: A Phase 2, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of VX-440 Combination Therapy in Subjects Aged 12 Years and Older With Cystic Fibrosis | | | | |
| I have read Protocol VX15-440-101, Version 2.0, and agree to conduct the study according to its terms. I understand that all information concerning VX-440, tezacaftor, and ivacaftor and this protocol supplied to me by Vertex Pharmaceuticals Incorporated (Vertex) is confidential. | | | | |
| Printed Name | | | | |
| Signature | | Dat | e | |